## **Study Identification**

Unique protocol identification number: STUDY00004627

Brief Title: Training LHD's to disseminate evidence-based interventions to small work sites

Official Training Local Health Departments to Disseminate Evidence-Based Interventions to Small and

Title: Low-Wage Worksites

Secondary 2R01CA160217 [U.S. NIH Grant/Contract Award Number]

IDs: NCI-2021-02876 [Registry ID: CTRP (Clinical Trial Reporting Program)]

RG1121453 [Fred Hutch/University of Washington Cancer Consortium]

Document date: September 24, 2019

The protocol for the randomized trial reviewed by the University of Washington Institutional Review Board appears below. Information about an additional study (Aim 1 activities in the protocol) outside of the randomized trial and information that describes individuals' names or intellectual property has been redacted.





## **INSTRUCTIONS**

- <u>If you are requesting a determination</u> about whether your activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example 1.1 must be answered.
- Answer all questions. If a question is not applicable to your research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- The word "you" refers to the researcher and all members of the research team, unless otherwise specified.
- For collaborative research, describe only the information that is relevant to you unless you are requesting that the UW IRB provide the review and oversight for your collaborators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to *Zipline*. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 Overview | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 Non-UW Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and Regulatory Issues |

## 1 OVERVIEW

**Study Title:** 

Disseminating Connect to Wellness Via Local Health Departments

1.1)Home institution. Identify the institution through which the lead researcher listed on the IRB application will conduct the research. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the POLICY: Use of the UW IRB.

University of Washington

1.2)Consultation history. Have you consulted with anyone at HSD about this study?

It is not necessary to obtain advance consultation. If you have: answering this question will help ensure that the IRB is aware of and considers the advice and guidance you were provided.



No

→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g. by email, phone call, in-person meeting).

We discussed this study with [redacted] via e-mail on 3/30/18 and 4/2/18, and via telephone on 8/21/2018. We also consulted with [redacted] via phone and e-mail in July/August 2019.

1.3) Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

The current IRB application is for a National Cancer Institute funded competing renewal of our HealthLinks R01 (grant number R01CA160217). The former proposal was to test the effectiveness of the HealthLinks intervention for small worksites. The IRB number was 45447EJ, study title: HealthLinks Trial: Increasing Implementation of Evidence-Based Interventions at Low-Wage Worksites, and the lead researcher was Margaret (Peggy) Hannon.

Please note that we changed the name of the intervention for the current project and IRB proposal. We learned that the name HealthLinks was trademarked by another group, and changed the name to Connect to Wellness. However, the intervention is the same.

Finally, the current IRB application is related to application number 00004627, which we submitted in April 2018 as part of our Just In Time package to NCI and modified for our initial study (Aim 1) in November 2018 and August 2019.

1.4) Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect your proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.



No

→ If yes, briefly describe the urgency or deadline as well as the reason for it.

1.5)Objectives Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If your application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

The primary goals of this study are to (a) scale up Connect to Wellness by training staff in local health departments across the United States to deliver Connect to Wellness to small worksites in their communities, and (b) conduct a trial comparing the effectiveness and costs of two different implementation strategies.

It has been previously proven that Connect to Wellness is effective. Our objective now is to determine the best way to implement it. Although the local health departments will be involved in collecting identifiable data, they are not engaged in the research because we are not testing the efficacy of Connect to Wellness.

Study goals will be achieved through three aims:

Aim 1: Conduct formative research (interviews and focus groups) with state and local health departments Aim 2: Test two different implementation strategies with local health departments: 1) standard Connect to Wellness training and technical assistance and 2) standard Connect to Wellness training plus enhanced technical assistance Aim 3: Measure the costs of each implementation strategy

**1.6) Study design**. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in assigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

Aim 1 activities are qualitative. We will conduct semi-structured interviews and focus groups with participants via online and telephone methods.

Aim 2 is a hybrid type III randomized controlled trial comparing two different Connect to Wellness implementation strategies. We will randomize 40 local health departments to receive either a 1) standard training and technical assistance or 2) standard training plus enhanced technical assistance.

Aim 3 will measure the costs associated with each implementation strategy via process measures (e.g. tracking worksheets) and conduct a cost analysis based on this data.

**1.7)Intent**. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.

| Descriptor |
|---|
| 1. Class project or other activity whose purpose is to provide an educational experience for the researcher (for example, to learn about the process or methods of doing research). |
| 2. Part of an institution, organization, or program's own internal operational monitoring. |
| 3. Improve the quality of service provided by a specific institution, organization, or program. |
| 4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that: |
| Are expected to be applicable to a larger population beyond the site of data collection or the specific subjects studied, or |
| <ul> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships,<br/>or to inform policy beyond the study.</li> </ul> |
| 5. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 6. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 7. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 8. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 9. Expanded access use of a drug or device not yet approved for this purpose |
| 10. Use of a Humanitarian Use Device |
| 11. Other. Explain: |

- **1.8 Background, experience, and preliminary work**. Answer this question <u>only</u> if your proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for your proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that your project is intended to address.

This should be a plain language description. Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

Cancer and other chronic diseases are the leading causes of death in the United States. Several preventable risk behaviors, including physical inactivity, unhealthy eating, missed cancer screenings, and tobacco use increase disease risk. Evidence-based interventions significantly reduce each of these risk behaviors. Most adults in the United States are employed, and worksites can implement evidence-based interventions to support worker health.

However, small worksites (businesses with less than 250 employees) infrequently implement these interventions and face budget, capacity, and partnership challenges in doing so. To assist these worksites, we previously partnered with the American Cancer Society to create and test *Connect to Wellness*, a program to disseminate evidence-based interventions and provide implementation support. The findings from this work show that *Connect to Wellness* is effective, but wider dissemination of this program has yet to occur.

Local health departments cover most communities, and most local health department goals include preventing chronic disease. Previous studies of local health department activities and investments show positive associations between their efforts and health outcomes in communities. Given this information, these departments have the potential to assist with the dissemination of *Connect to Wellness* nationwide. While local health departments are a vital part of community-based chronic disease practice, they are underrepresented in implementation research.

**b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you or your team have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: You have already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study you are now proposing to do; you have already done a small pilot study showing that the reading skills intervention you plan to use is feasible in an after-school program with classroom aides; you have experience with the type of surgery that is required to implant the study device; you have a study coordinator who is experienced in working with subjects who have significant cognitive impairment.

We previously tested the *Connect to Wellness* intervention in a pilot study and randomized controlled trial. In 2012, we trained a health educator in a rural local health department to deliver *Connect to Wellness*. Training included in-person meetings and observations. To make training and technical assistance more sustainable, we

developed and pilot-tested a distance-training model with success in several local health departments in Washington State.

**1.9 Supplements**. Check all boxes that apply, to identify Supplements you should complete and upload to the **Supporting Documents** SmartForm in **Zipline**.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Defense |
| | <b>Department of Energy</b> The research involves Department of Energy funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Energy |
| | <b>Drug, biologic, botanical, supplement</b> Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of your research | ZIPLINE SUPPLEMENT: Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | ZIPLINE SUPPLEMENT: Exception from Informed Consent for Emergency Research (EFIC) |
| | Genomic data sharing Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other researchers, and you are asking the UW to provide the required certification or to ensure that the consent forms can be certified | ZIPLINE SUPPLEMENT:<br>Genomic Data Sharing |
| | <b>Medical device</b> Procedures involve the use of <u>any</u> medical device, even if the device is not the focus of your research, except when the device is FDA-approved and is being used through a clinical facility in the manner for which it is approved | ZIPLINE SUPPLEMENT: Devices |
| | Multi-site study (You are asking the UW IRB to review one or more sites in a multi-site study.) | ZIPLINE SUPPLEMENT: Participating Site in Multi- Site Research |
| | Participant results sharing Individual research results will be shared with subjects. | ZIPLINE SUPPLEMENT: Participant Results Sharing |
| х | None of the above | |

# **2 PARTICIPANTS**

| <b>2.1</b> Participants. Describe the general characteristics of the subject populations or groups, including age range, gender, health status, and any other relevant characteristics. |
|---|
| Aim 1: [redacted] |
| Aims 2/3: The first group of participants will be <u>local health department staff</u> , coming from 40 local health departments across the U.S., who will be trained to recruit and deliver Connect to Wellness to small worksites in their communities. The second group of participants will be <u>representatives from these worksites</u> , who will provide feedback about their experiences with Connect to Wellness via a brief satisfaction survey. To conduct the cost analysis for Aim 3, we will use data collected by members of the research team and by local health department staff. |
| (2.2) Inclusion and exclusion criteria. |
| a. Inclusion criteria. Describe the specific criteria you will use to decide who will be included in your study from among interested or potential subjects. Define any technical terms in lay language. |
| Aim 1: [redacted] |
| Aims 2/3: Local health departments in the 50 states and District of Columbia will be eligible to participate in the randomized controlled trial. Additional eligibility criteria include willingness to support one or more staff members to participate in <i>Connect to Wellness</i> training and the project for two years, and to have these staff recruit 15 or more worksites for <i>Connect to Wellness</i> over 24 months. We will recommend to local health department staff that they focus on recruiting worksites with 20-200 employees (i.e. worksites with fewer resources for workplace health promotion, and for which the strongest evidence for the effectiveness of <i>Connect to Wellness</i> is present). The worksite representatives will need to be able to speak and read English, and be knowledgeable about health and wellness at the worksite (e.g. HR manager). We expect that representatives will be at least 18 years of age or older. |
| b. Exclusion criteria. Describe the specific criteria you will use to decide who will be excluded from your study from subjects who meet the inclusion criteria listed above. Define any technical terms in lay language. |
| Aim 1: [redacted] |
| Aims 2/3: Local health departments who are not able to support staff to participate in <i>Connect to Wellness</i> will be excluded from the study. |
| 2.3 Prisoners. IRB approval is required in order to include prisoners in research, even when prisoners are not an intended target population. |
| a. Will you recruit or obtain data from individuals that you know to be prisoners? |
| For records reviews: if the records do not indicate prisoner status and prisoners are not a target population, select "No". See the <u>WORKSHEET: Prisoners</u> for the definition of "prisoner". |
| x No Yes → If yes, answer the following questions (i – iv). |
| i. Describe the type of prisoners, and which prisons/jails: |

| living conditions, medical care, qual | h is whether the effect of participation on prisoners' general ity of food, amenities, and opportunity for earnings in prison ifficult for prisoners to adequately consider the research risks. nces of this? |
|---|---|
| | sure that (a) your recruitment and subject selection procedures nd (b) prison authorities or other prisoners will not be able to ular prisoners from participating. |
| Washington State: check the box be or facilitate the use of a prisoner's p | rs in federal facilities or in state/local facilities outside of elow to provide your assurance that you will (a) not encourage participation in the research to influence parole decisions, and edvance (for example, in a consent form) that participation in his or her parole. |
| Confirmed | |
| <b>b.</b> Is your research likely to have subjects who become | prisoners while participating in your study? |
| For example, a longitudinal study of youth with drug pr point during the study. | oblems is likely to have subjects who will be prisoners at some |
| procedures and/or data collection w | er while participating in your study, will you continue the study while the subject is a prisoner? Occedures and/or data collection you will continue with prisoner |
| any of these populations that you will purposefully include population is an inclusion criterion for your study.) | ise of the subject populations listed here. Check the boxes for de in your research. (In other words, being a part of the |
| The WORKSHEETS describe the criteria for approval but do i | not need to be completed and should not be submitted. |
| Population | Worksheet |
| Fetuses in utero | WORKSHEET: Pregnant Women |
| Neonates of uncertain viability | WORKSHEET: Neonates |
| Non-viable neonates | WORKSHEET: Neonates |
| Pregnant women | WORKSHEET: Pregnant Women |

| | non U.S. indigenous populations. Will you actively recruit from Native American or non-U.S. ons through a tribe, tribe-focused organization, or similar community-based organization? |
|---|---|
| | e defined in international or national legislation as having a set of specific rights based on their historica<br>Pritory and their cultural or historical distinctiveness from other populations that are often politically |
| Examples: a reservat | ion school or health clinic; recruiting during a tribal community gathering |
| x No | |
| | , name the tribe, tribal-focused organization, or similar community based organization. The UW IF<br>cts that you will obtain tribal/indigenous approval before beginning your research. |
| САВС | and that you thin obtain thou, margemous approval service segmining your research |
| 'hind vantu avlaiasta | Will you called write identifiable information about ather individuals from your subjects? |
| | Will you collect private identifiable information about other individuals from your subjects? nclude: collecting medical history information or contact information about family members, |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest | |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest | nclude: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest readily identify the grown of the composition of the | nclude: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you and parents, then you are not collecting private identifiable information about the grandparents. es, these individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you andparents, then you are not collecting private identifiable information about the grandparents. These individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you and parents, then you are not collecting private identifiable information about the grandparents. es, these individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest readily identify the grown of the composition of the | nclude: collecting medical history information or contact information any direct or indirect identifier that, alone or in combination, would alloudily identify the person. For example, suppose that you are studying imnions about their grandparents but you do not obtain names or other information and parents, then you are not collecting private identifiable information es, these individuals are considered human subjects in your study. D |

# **2.7 Number of subjects.** Can you predict or describe the maximum number of subjects (or subject units) you need to complete your study, for each subject group?

<u>Subject units</u> mean units within a group. For most research studies, a group will consist of individuals. However, the unit of interest in some research is not the individual. Examples:

- Dyads such as caregiver-and-Alzheimer's patient, or parent and child
- Families
- Other units, such as student-parent-teacher

<u>Subject group</u> means categories of subjects that are meaningful for your research. Some research has only one subject group – for example, all UW students taking Introductory Psychology. Some common ways in which subjects are grouped include:

- By intervention for example, an intervention group and a control group.
- By subject population or setting for example, urban versus rural families
- By age for example, children who are 6, 10, or 14 years old.

The IRB reviews the number of subjects you plan to study in the context of risks and benefits. You may submit a Modification to increase this number at any time after you receive IRB approval. If the IRB determines that your research involves no more than minimal risk: you may exceed the approved number and it will not be considered non-compliance. If your research involves more than minimal risk: exceeding the approved number will be considered non-compliance.



→ If no, provide your rationale in the box below. Also, provide any information you can about the scope/size of the research. You do not need to complete the table.

Example: you may not be able to predict the number of subjects who will complete an online survey advertised through Craigslist, but you can state that you will post your survey for two weeks and the number who respond is the number who will be in your study.



→ If yes, for each subject group, use the table below to provide your estimate of the maximum desired number of individuals (or other subject unit, such as families) who will complete the research.

| or clinical trials: provide numbers for your site and for estudy-wide total number |
|---|
| 5 |
| ) |
| ) |
| )-80 |
| 00 |
| 5 |

# **3 NON-UW RESEARCH SETTING**

# Complete this section only if your research will take place outside of UW and Harborview

| Intext. Culturally-appropriate procedures and an understanding of local context are an important part of ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. Ses: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male their; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. Secific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: Secific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: Secific laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. Secific laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. Seally authorized representative — laws about who can serve as a legally authorized representative (and we spriority when more than one person is available) vary across states and countries. |
|---|
| ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. es: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male her; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. eral site maintains an international list of human research standards and requirements: www.hhs.gov/ohrp/international/index.html ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. eally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. es: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male her; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. eral site maintains an international list of human research standards and requirements: www.hhs.gov/ohrp/international/index.html ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. eally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ther; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. The property of a group. The property of the maintains an international list of human research standards and requirements: The property of the provide consent vary ross states, and across countries. The property of the provide consent vary ross states, and across countries. The property of the proper |
| ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary oss states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary oss states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and w |
| e of healthcare records – many states (including Washington State) have laws that are similar to the deral HIPAA law but that have additional requirements. |
| ecific administrative or ethical requirements. Describe local administrative or ethical requirements that affect search. |
| e: A school district may require you to obtain permission from the head district office as well as school principals befo<br>ching teachers or students; a factory in China may allow you to interview factory workers but not allow you to pay |
| e :: |

**4.1** Recruiting and Screening. Describe how you will identify, recruit, and screen subjects. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

# Aim 1: [redacted]

#### Aims 2/3:

To recruit local health departments for the trial, The National Association for Chronic Disease Directors will include us on the agenda for a webinar or in-person meeting of the state chronic disease directors. To ensure outreach to the entire group, follow-up email communication will go to the state-level voting members. At the meeting, we will present *Connect to Wellness* and its evidence-base and describe the proposed trial. We will request that state chronic disease directors share this information with their local health departments, and will offer to follow-up individually if they have questions or concerns. We will work the state chronic disease directors who believe one or more local health departments in their state would be interested in the study to identify the best ways to recruit these local health departments. The state chronic disease director may make a referral to the local health department, linking their director or appropriate staff to the research team, or s/he may prefer to send out recruitment materials to local health department directors directly. If this approach does not yield 40 local health departments, we may use one or more of the following strategies to reach local health department directors directly: The director of the UW's Public Health Training Center, the Northwest Center for Public Health Practice, is a co-investigator for this study and is able to refer us to local health department directors in the multi-state region served by her Center. We may also advertise the study through the National Association of City and County Health Officials and/or through the Association of State and Territorial Health Officials (email blast or newsletter).

Recruitment materials will direct local health department directors or staff to contact a member of our research team via telephone for more information. Local health departments who contact us will be given more information about the study so that they understand the project purpose and duration, requirements of staff time, recruitment expectations, and data requirements. This conversation will serve as part of the screening process, whereby local health departments who cannot dedicate the staff and time to this project will not be invited to participate in the trial.

To recruit worksite representatives for the brief satisfaction survey, we will generate a random sample of five worksites per local health department (e.g. via a random numbers table) and contact representatives by e-mail or telephone to schedule a time to complete the brief satisfaction survey.

### 4.2 Recruitment materials.

a. What materials (if any) will you use to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

#### Aim 1:

[redacted]

### Aims 2/3:

We will have presentation materials (e.g. PowerPoint, talking points, and notes) to do initial outreach with state chronic disease directors. We will use written materials and a telephone script to talk to interested local health departments about the study. The content of the written materials will also reside on a website about *Connect to Wellness* for the recruitment phase.

b. Upload descriptions of each type of material (or the materials themselves) to the Consent Forms and Recruitment Materials SmartForm of **Zipline**. If you will send letters to the subjects, the letter should include a statement about how you obtained the subject's name, contact information, and any other subject-specific information (such as a health condition) that is mentioned in the letter.

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- You could provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, you might include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). In doing so, you would not need to submit a Modification if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, you might state that the flyer will list one or a few of the major inclusion/exclusion
- For the description of a video or a website, you might include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).
- 4.3 Relationship with participant population. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



No

→ If yes, describe the nature of the relationship.

[redacted] at the National Association of Chronic Disease Directors (a co-investigator on the grant) consults with state-level public health leaders to improve their organization's practices. [redacted] (also a co-investigator on this grant) works for the Northwest Center for Public Health Practice, which provides training to local health departments. Neither manage or have direct oversight of individuals working in these settings.

- **4.4 Payment to participants**. Describe any payment you will provide, including:
  - The total amount/value
  - Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include information about the number and amount of payments, and especially the time when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Do not include a description of any expenses that will be reimbursed.

| N I | / A |
|-----|-------------------|
| 1/1 | <i>,</i> $\Delta$ |

| | stude | nts; a | tary compensation. Describe any non-monetary compensation you will provide. Example: extra credit for toy for a child. If you will be offering class credit to students, you must provide (and describe) an alternate students to earn the extra credit without participating in your research. |
|---|---|---|---|
| | N/A | | |
| 4.6 | Will y | ou ac | cess or obtain data or specimens for recruiting and screening procedures prior to enrollment? |
| | | ionnai | ames and contact information; the information gathered from records that were screened; results of screening res or screening blood tests; Protected Health Information (PHI) from screening medical records to identify possible |
| | | No | → If no, skip the rest of this section; go to question 5.1. |
| | х | Yes | → If yes, describe any data and/or specimens (including PHI) you will access or obtain for recruiting and screening and whether you will retain it as part of the study data. |
| | | | Aim 1:<br>[redacted] |
| | | | Aims 2/3: We may obtain the names and contact information for individuals within the local health departments from the state chronic disease directors, should the director provide a referral for us. |
| 4.7 | | | r recruiting and screening. Will you obtain consent for any of the recruiting and screening procedures? Consent of Adults asks about consent for the main study procedures). |
| | | | ncludes: consent from individuals for their own participation; parental permission; assent from children; consent<br>Ily authorized representative for adult individuals who are unable to provide consent. |
| | •<br>•<br>• | Foi<br>fro<br>Foi<br>Foi | r a study in which names and contact information will be obtained from a registry: the registry should have consent m the registry participants to release their names and contact information to researchers. r a study in which possible subjects are identified by screening records: there will be no consent process. r a study in which individuals respond to an announcement and call into a study phone line: the study team person king to the individual may obtain non-written consent to ask eligibility questions over the phone. |
| | х | No<br>Yes | <ul> <li>→ If no, skip the rest of this section; go to <u>question 5.1</u>.</li> <li>→ If yes, describe the consent process.</li> </ul> |
| | | | in yes, describe the sonsent processi |
| | | | <ul> <li>a. <u>Documentation of consent</u>. Will you obtain a written or verifiable electronic signature from the subject on a consent form to document consent for all of the <u>recruiting and screening procedures</u>?</li> <li>→ If no, describe the information you will provide during the consent process and for</li> </ul> |
| | | | No which procedures. |
| | | | Yes → If yes, upload the consent form to the <b>Consent Forms and Recruitment Materials</b> page of <b>Zipline</b> . |

## **5 PROCEDURES**

5.1 Study procedures. Using lay language, provide a complete description of the study procedures, including the sequence, intervention or manipulation (if any), drug dosing information (if any), use of records, time required, and setting/location. If it is available and you think it would be helpful to the IRB: Upload a study flow sheet or table to the Supporting Documents SmartForm in *Zipline*.

For studies comparing standards of care: It is important to accurately identify the research procedures. See UW IRB <u>POLICY:</u>
<u>Risks of Harm from Standard Care</u> and the draft guidance from the federal Office of Human Research Protections, <u>"Guidance on Disclosing Reasonably Foreseeable Risks in Research Evaluating Standards of Care"; October 20, 2014.</u>

# Aim 1: [redacted]

#### Aim 2:

Once a local health department has been recruited to participate in the study, they will be randomized to one of two conditions for the trial: 1) standard training and technical assistance or 2) standard training plus enhanced technical assistance.

Briefly, local health department staff will be trained to deliver the *Connect to Wellness* intervention to worksites that they recruit. In the Assessment phase, staff will measure current worksite implementation of physical activity, nutrition, cancer screening, and tobacco cessation evidence-based interventions (with the Baseline Employer Assessment Survey). [redacted] During the Implementation phase (months 3-12), the worksite begins adopting the recommended evidence-based intervention policies and programs and promoting them to workers. At the conclusion of the Implementation phase (month 12), the local health department staff will re-administer the Employer Assessment Survey. After this 12-month period, worksites are able to contact the local health department for technical assistance; the health department may also periodically contact worksites with study updates or to provide relevant materials or offer implementation support.

Once a local health department is assigned to the standard arm, a member of the research team will contact staff to arrange dates for the training sessions, ship materials for the worksites (e.g. toolkits), and provide a detailed *Connect to Wellness* protocol to use with worksites that they recruit. The research team will e-mail information about the *Connect to Wellness* training website and ensure that staff are able to register. Local health department staff will attend three online training webinars, each lasting two hours, in groups of five. (Note: Five refers to the number of local health departments represented in each group). These real-time webinars will be supported by Zoom software. Topics covered in this training will include an introduction to *Connect to Wellness*, methods for recruiting worksites, how to administer the Employer Assessment Survey, how to create and deliver the recommendations report, an overview of intervention implementation and programming, how to track (e.g. their interactions with worksites, time spent on project), and discussion of common barriers and solutions. At the conclusion of the third training webinar, we will work with each group of local health departments to identify a time for monthly group technical assistance calls, where staff will have time to share lessons learned and success stories. Features will be added to the *Connect to Wellness* website to encourage communication between members of each five-local health department group, such as discussion forums and instant chat.

Local health departments assigned to the enhanced arm will undergo initial and online training procedures as described above. Each group will also have a monthly technical assistance call and access to the online peer-communication tools described above. In addition, local health departments in this arm will have one-on-one telephone access to a member of our research team. They can call her for advice; she will proactively contact each local health department in this arm monthly if they have not contacted her during that time. Enhanced support will be given for 24 months, the same length as the study period for this aim.

Throughout the study period, members of the research team will contact local health department staff via e-mail or telephone to obtain study data (measures described in Section 5.2). REDCap will be primarily used for data collection. Local health department staff will provide members of the research team with the contact information of worksite representatives from a sample of the worksites they recruit and deliver Connect to Wellness to. These representatives will be contacted via e-mail or telephone to schedule a time to complete the brief satisfaction survey. The survey will be administered by telephone.

#### Aim 3:

Following methods recommended by previous studies, we will assess the overall costs to implement the standard and enhanced training and technical assistance strategies, including all training and technical assistance activities conducted by the research team as well as activities performed by local health departments.

(5.2) Data variables. Describe the specific data you will obtain (including a description of the most sensitive items). If you would prefer, you may upload a list of the data variables to the **Supporting Documents** SmartForm instead of describing the variables below.

# Aim 1: [redacted]

#### Aims 2/3:

We will collect the following data from local health department staff: 1) <u>local health department characteristics</u>; 2) <u>satisfaction with training and technical assistance</u>; 3) <u>implementation and intent to maintain *Connect to Wellness*</u>; and 5) <u>staff and worksite activities</u>, which will help us to determine which implementation strategy is more effective and the costs associated with each implementation strategy.

- 1. We will measure local health department characteristics using items from the 2016 National Profile of Local Health Departments. Sample measures include state, population size served, geographic region served, and governance (state, local, or shared). A co-investigator on this grant will pull these measures from the 2016 National Profile data, and we will ask staff to confirm their local health department's information.
- 2. We will ask staff to complete a brief online evaluation to assess satisfaction with and understanding of the training. We will also ask them to complete a satisfaction survey with the *Connect to Wellness* technical assistance they receive every six months and ask staff in the enhanced arm about their satisfaction with one-on-one support.
- 3. We will adapt adoption, implementation, and maintenance items from the Prevention Program Assessment and ask local health department staff to complete these items at 12 and 24 months to assess their implementation and intent to maintain *Connect to Wellness*. The Program Sustainability Assessment Tool will be used as an additional measure to assess capacity to maintain *Connect to Wellness*.
- 4. Staff will be asked to track and provide data on the following: number of meetings, phone contacts, and emails with each worksite; number of worksites that complete *Connect to Wellness*; and personnel time, travel costs, and costs for printing materials for worksites.

In addition to the measures described above, local health department staff will provide us with the Employer Assessment Survey data that they collect from the worksites, which will further help us to determine which implementation strategy is more effective. The identities of the worksite representatives that we ask to complete the brief satisfaction survey will be known to us for recruitment purposes, but we will not retain this information as part of our study data. The identities of these representatives will not be known otherwise. For the employer assessment survey, we will only know the worksite name and corresponding ID number.

Lastly, the research team will track local health department's participation in *Connect to Wellness* training sessions and their attendance at technical assistance calls (group calls and one-on-one calls). The *Connect to Wellness* training and support website will track each local health department's log-ins, visits to the website, and material downloads.

For the worksite representatives, we will collect data on their satisfaction with Connect to Wellness.

**5.3** Data sources. For all types of data that you will access or collect for this research: Identify whether you are obtaining the data from the subjects (or subjects' specimens) or whether you are obtaining the data from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

### Aim 1:

[redacted]

Aims 2/3:

The data described above will come from members of the research team, local health department staff, and worksite representatives.

(5.4) Retrospective/prospective. For all types of data and specimens that you will access or collect for this research: do all data and specimens to be used in the research exist (for example, in subjects' medical records) at the time this application is being submitted for initial review?



No Yes

Include any necessary comments or explanation below (Note that for most studies this can be left blank):

**5.5 Identifiability of data and specimens**. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and to assist you in identifying relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain". Identifiable means that the identity of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

**Direct identifiers** are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of your data that is (when taken together) identifiable.

**Indirect identifiers** are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

**Key** refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked to the codes.

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from **accessing**, which means to view or perceive data.

a. Will you or any members of your team have access to any direct or indirect identifiers?

| x |
|---|
|---|

Yes

→ If yes, describe which identifiers and for which data/specimens.

Aim 1: [redacted]

Aims 2/3:

| _ | We will know the names and contact information of local health department staff and worksite representatives. Electronic data files will refer to all worksites and local health departments via a numerical ID rather than by name. |
|---|---|
| No | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |
| <b>b.</b> Will you obtain | ain any direct or indirect identifiers? |
| x Yes | → If yes, describe which identifiers and for which data/specimens. |
| | We have to obtain names and contact information for recruitment and scheduling purposes. |
| No | → If no, select the reason(s) why you (and all members of your team) will not obtain direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |

| c. If you obtain any identifiers, indicate how the identifiers will be stored (and for which data). NOTE: Do not describe your data security plan here – we will ask for that information in section 9.6. |
|---|
| You will store the identifiers with the data. Describe the data to which this applies: |
| You will store identifiers and study data separately but you will maintain a link between the identifiers and the study data (for example, through the use of a code). Describe the data to which this applies: |
| For Aim 1[redacted] |
| We will use ID numbers to link study data with participant and organization (local health department and worksite) names. The file containing these ID numbers will be stored in a separate location. This applies to all data. |
| You will store identifiers separately from the study data, with no link between the identifiers and the study data. Describe the data to which this applies: |
| d. Research collaboration. Will individuals who provide you with coded information or specimens for your research also collaborate on other activities for this research? If yes, identify the activities and provide the name of the collaborator's institution/organization. Examples include but are not limited to: (1) study, interpretation, or analysis of the data that results from the coded information or specimens; and (2) authorship on presentations or manuscripts related to this work. |
| We do not anticipate sharing data with anyone outside the study team. |
| Newborn dried blood spots. Will you use newborn dried bloodspots collected in the United States on or after March 18, 2015? |
| Yes → If yes, is this research supported by any federal funding (including any fellowship or career development award that provides salary support)? |
| Yes → If yes, describe how you will ensure that the bloodspots were collected with parental permission (in compliance with a 2015 law that applies to federal-funded research). |
| Protected Health Information (PHI). Will you access, obtain, use, or disclose a participant's identifiable PHI for any leason (for example, to identify or screen potential subjects, to obtain study data or specimens, for study follow-up) what does not involve the creation or obtaining of a Limited Data Set? |
| PHI is individually-identifiable healthcare record information or clinical specimens from an organization considered a "covered entity" by federal HIPAA regulations, in any form or media, whether electronic, paper, or oral. <b>If you will use UW Medical Records, you must answer yes to this question.</b> |
| x No → If no, skip the rest of this question; go to question 5.8 |
| Yes → If yes, answer all of the questions below. |

| <b>a.</b> Describe the PHI you will access or obtain, and the reason for obtaining it. <i>Be specific</i> . |
|---|
| <b>b.</b> Is any of the PHI located in Washington State? |
| No<br>Yes |
| c. Describe how you will access or obtain the PHI. Be specific. |
| d. For which PHI will you obtain HIPAA authorization from the subjects by having them sign a HIPAA<br>Authorization form, before obtaining and using the PHI? |
| Confirm by checking the box that you will use the UW Medicine HIPAA Authorization form maintained on the HSD website if you will access, obtain, use, or disclose UW Medicine PHI. |
| Confirmed |
| e. For which PHI will you NOT obtain HIPAA authorization from the subjects? |
| Provide the following assurances by checking the boxes. |
| The PHI will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other research for which the use or disclosure of PHI would be permitted. |
| You will fulfill the HIPAA "accounting for disclosures" requirement. See <a href="UW Medicine Privacy">UW Medicine Privacy</a> <a href="Policy#25">Policy #25</a> . THIS IS ONLY FOR UW RECORDS. |
| There will be reasonable safeguards to protect against identifying, directly or indirectly, any patient in any report of the research. |
| 6.8 Genomic data sharing. Will you obtain or generate genomic data (as defined at http://osp.od.nih.gov/scientific-sharing/genomic-data-sharing-faqs/)? |
| x No |
| Yes $\rightarrow$ If yes, answer the question below. |
| a. Do you plan to send genomic data from this research to a national database (for example, NIH's dbGaP database)? |
| No Yes → If yes, complete the <u>ZIPLINE SUPPLEMENT Genomic Data Sharing</u> and upload it to the <b>Supporting Documents</b> SmartForm of <b>Zipline</b> . |

| <b>5.9 Whole genome sequencing.</b> For research involving biospecimens: Will the research include whole genome sequencing? | |
|---|---|
| Whole genome sequencing is sequencing of a human germline or somatic specimen with the intent to generate the genome exome sequence of that specimen. No Yes | e or |
| 5.10 Data and specimen sharing/banking. Are you likely to share some or all of the data, specimens, or subject contact information with other researchers or a repository/database for research purposes not related to this study, or to be them for your own future unspecified research uses? You are strongly encouraged to consider the broadest possible future plans you might have, and whether you will obtain consent now from the subjects for future sharing or unspecified uses. Answer YES even if you will only share information without identifiers. Answer NO if you are unlike to do any sharing, or if your only sharing will be through the NIH Genomic Data Sharing described in question 5.8. | le |
| data sharing as a condition of publication. "Sharing" may include: informal arrangements to share your banked data/specimens with other investigators; establishing a repository from which you formally share with others through writ | data/specimens with other investigators; establishing a repository from which you formally share with others through written agreements; or sending your data/specimens to a third party repository/archive/entity such as the Social Science Open Access |
| x No Yes → If yes, answer all of the questions below. | |
| <ul> <li>a. Describe <u>what will be stored</u>, including whether any direct or indirect (e.g., subject codes) identified will be stored.</li> </ul> | |
| <b>b.</b> Describe <u>what will be shared</u> , including whether direct identifiers will be shared and (for specime what data will be released with the specimens. | ns) |
| c. Who will oversee and/or manage the sharing? | |
| d. Describe the possible future uses, including limitations or restrictions (if any) on future uses of users. As stated above, consider the broadest possible uses. Examples: data will be used only for cardiovascular research; data will not be used for research on population origins. | r |
| e. Consent. Will you obtain consent now from subjects for the banking and/or future sharing? No Yes → If yes, be sure to include the information about this consent process in the consent form (if there is one) and in your answers to the consent questions in Section 8. | ent |

| Yes → If yes, describe how, and whether there are any limitations | on withdrawal |
|---|---|
| Example: data can be withdrawn from the repository but can are released. | |
| g. Agreements for sharing or release. Confirm by checking the box that you (and, if applicable, UW Medicine) policies that require a formal agreeme the recipient for release of data or specimens to individuals or entities or databases. | nt between you and |
| Data Use Agreements or Gatekeeping forms are used for data; Material Transfe<br>for specimens (or specimens plus data. Do not attach your template agreement<br>reviews nor approves them | _ |
| Confirmed | |
| <b>5.11 Communication with subjects during the study</b> . Describe the types of communication (if any) already-enrolled subjects during the study. Provide a description instead of the actual material | • |
| Examples: email, texts, phone, or letter reminders about appointments or about returning study mat questionnaire; requests to confirm contact information. | erials such as a |
| Aim 1: [redacted] | |
| Aims 2/3: | |
| Research team members will have multiple types of contact with the local health department phone calls, and in-person meetings. Research team members' only direct contact with works be to collect their brief satisfaction survey data once, after the worksite has been doing Conne months. | te representatives will |
| <b>5.12 Future contact with subjects</b> . Do you plan to retain any contact information you obtain for you can be contacted in the future? | ır subjects so that they |
| No Yes → If yes, describe the purpose of the future contact, and whether use of the contact limited to your team; if not, describe who else could be provided with the contact Describe your criteria for approving requests for the information. | |
| Examples: inform subjects about other studies; ask subjects for additional information access that is not currently part of the study proposed in this application; obtain and | |
| Aim 1: [redacted] | |
| Aims 2/3: | |

f. Withdrawal. Will subjects be able to withdraw their data/specimens from banking or sharing?

not be retained after the study closes.

The contact information for subjects (local health department staff and worksite representatives) will

# **5.13 Alternatives to participation.** Are there any alternative procedures or treatments that might be advantageous to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.

| х | No |
|---|----|
| | Va |

→ If yes, describe the alternatives.

- **5.14 Upload to the Supporting Documents** SmartForm of *Zipline* all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points you will use to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records, or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - NOTE: Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics you will cover and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.
  - For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those interactions. If this applies to your research, provide a description of the process by which you will establish the data collection/questions as you interact with subjects, how you will document your data collection/questions, the topics you plan to address, the most sensitive type of information you will plan to gather, and the limitations (if any) on topics you will raise or pursue.

### Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process you will use for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which you are seeking general approval. (See the **NOTE** bullet point in the instructions above.)

| Aim 1: |
|-----------|
| [redacted |

**5.15 Send HSD** a <u>Confidentiality Agreement</u> if you will obtain or use any private identifiable UW records without subject's written consent (for example, screening medical records or class grades to identify possible subjects).

The Confidentiality Agreement form must be completed, printed, signed, and mailed to the Human Subjects Division at Box 359470. Your IRB application cannot be approved until we receive the Confidentiality Agreement.

# 6 CHILDREN (MINORS) and PARENTAL PERMISSION

**(6.1)Involvement of minors.** Does your research include minors (children)?

**Minor or child** means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State.
- The generic age of consent may be different in other states, and in other countries.

| × | No<br>Yes | → If no, go to Section 8. | | |
|---|---|---|---|---|
| | | → If yes, provide the age range of the minor subjects for this study and the legal age for population(s). If there is more than one answer, explain. | consent ii | ı your |
| | Don't | <ul> <li>→ This means is it not possible to know the age of your subjects. For example, some research involving social media, the Internet, or a dataset that you obtaresearcher or from a government agency. Go to <a href="Section 8">Section 8</a>.</li> </ul> | | |
| as<br>the | "passive"<br>ey have b | rmission. Parental permission means actively obtaining the permission of the parents. The or "opt out" permission where it is assumed that parents are allowing their children to peen provided with information about the research and have not objected or returned a father children to participate. | articipate | because |
| a. | Will you o | obtain parental permission for: | | |
| | All of | your research procedures $\rightarrow$ Go to <u>question 6.2b.</u> | | |
| | None | of your research procedures Use the table below to provide your justification, 6.2b. | and skip o | uestion |
| | Some | of your research procedures Use the table below to identify the procedures for not obtain written parental permission. | or which yo | ou will |
| | | onsider all research procedures and plans, including screening, future contact, and sharing/bai<br>or future work. | nking of da | ta and |
| Describe the procedures or Children data/specimen collection (if any) for Group <sup>1</sup> which there will be NO parental permission <sup>2</sup> | | data/specimen collection (if any) for | Will you<br>them ab<br>resea | out the |
| | | | YES | NO |

| | | | — |
|---|---|---|---|
| | | Ш | |
| Tak | ble footnotes | | |
| 1. | If your answer is the same for all children groups or all procedures, you can collapse your answer across the procedures. | e groups an | d/or |
| 2. | If you plan to obtain identifiable information or biospecimens without parent permission, any waiver grant not override parents' refusal to provide broad consent (for example, through the Northwest Biotrust). | - | RB does |
| 3. | Will you inform them about the research beforehand even though you are not obtaining active permission? | | |
| | <b>b.</b> Indicate by checking the appropriate box(es) your plan for obtaining parental permission | | |
| | Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably availating one parent has legal responsibility for the care and custody of the child | ble; or wh | en only |
| | One parent, even if the other parent is alive, known, competent, reasonably available, and share responsibility for the care and custody of the child. | ares legal | |
| | This is all that is required for minimal risk research. | | |
| | If you checked both boxes, explain: | | |
| 6.3 | <b>B Children who are wards.</b> Will any of the children be wards of the State or any other agency, institutio | n, or entity | <b>'</b> ? |
| | No | | |
| | Yes If yes, an advocate may need to be appointed for each child who is a ward. The advocate addition to any other individual acting on behalf of the child as guardian or in loco par individual can serve as advocate for all children who are wards. | | |
| | Describe who will be the advocate(s). Your answer must address the following point: • Background and experience | 5: | |
| | <ul> <li>Willingness to act in the best interests of the child for the duration of the re</li> <li>Independence of the research, research team, and any guardian organization</li> </ul> | | |

# 7 ASSENT OF CHILDREN (MINORS)

Go to <u>Section 8</u> if your research does not involve children (minors).

**7.1 Assent of children (minors)**. Though children do not have the legal capacity to "consent" to participate in research, they should be involved in the process if they are able to "assent" by having a study explained to them and/or by reading a simple form about the study, and then giving their verbal choice about whether they want to participate. They may also provide a written assent if they are older. See **WORKSHEET: Children** for circumstances in which a child's assent may be unnecessary or inappropriate.

| All of your research | n procedures and child groups | → Go to question <b>7.2.</b> |
|---|---|---|
| None of your resea | arch procedures and child groups | → Use the table below to provide your justification, then skip to question 7.5. |
| Some of your resea | arch procedures and child groups | → Use the table below to identify the procedures for which you will not obtain assent. |
| Be sure to consider all resea<br>specimens for future work. | arch procedures and plans, including screen | ing, future contact, and sharing/banking of data and |
| Children Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which assent will NOT be obtained | Reason why you will not obtain assent |
| | for all children groups or all procedures, you | u can collapse your answer across the groups and/or |
| procedures. | | |
| ages, answer separately fo | • | group. If your research involves children of different glish speakers, include a description of how you will |
| ages, answer separately fo | or each group. If the children are non-Eng | <del>-</del> |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description | or each group. If the children are non-Englend the information you provide. | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Desiverbal indications) during | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object the research, and what you will do in res | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description of assent. 7.4 Documentation of assent. assent? | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object the research, and what you will do in res | glish speakers, include a description of how you will cition or resistance to participation (including non-sponse. |
| ages, answer separately for ensure that they comprehence. 7.3 Dissent or resistance. Deserverbal indications) during 7.4 Documentation of assent. assent? None of your research. | or each group. If the children are non-Engiend the information you provide. cribe how you will identify a child's object the research, and what you will do in research. | glish speakers, include a description of how you will ction or resistance to participation (including non-sponse. ribes whether you will obtain documentation of → Use the table below to provide your |

| | Children | Describe the procedures or data/specimen collection (if any) for which assent |
|---|---|---|
| | Group <sup>1</sup> | will NOT be documented |
| | · | |
| Table | footnotes | |
| 1. If | | ne for all children groups or all procedures, you can collapse your answer across the groups and/or |
| ć | a. Describe how you value a description of wh | will document assent. If the children are functionally illiterate or are not fluent in English, include nat you will do. |
| CI<br>OI<br>OI<br>SU | the information she in Word, if possible hildren who reach the hildren who were enrotain it for the first time hildren who reach the higoing interactions or object's identify is rea | ine. Assent materials are not required to provide all of the standard elements of adult consent; ould be appropriate to the age, population, and research procedures. The documents should be elements age of consent during participation in longitudinal research. Olled at a young age and continue for many years: It is best practice to re-obtain assent (or to me, if you did not at the beginning of their participation). Elegal age of consent: You must obtain informed consent from the now-adult subject for (1) any interventions with the subjects, or (2) the continued analysis of specimens or data for which the dily identifiable to the researcher, unless the IRB waives this requirement. |
| 1 | <ul> <li>If you plan to contact.</li> </ul> | s (if any) to obtain consent for children who reach the legal age of consent. obtain consent, describe what you will do about now-adult subjects whom you are unable to plan to obtain consent or think that you will be unable to do so, explain why. |
| | | rements. (This is for your information only; no answer or response is required.) Researchers are ining whether their research conducted in schools, with student records, or over the Internet |

- comply with permission, consent, and inspection requirements of the following federal regulations:
  - PPRA Protection of Pupil Rights Amendment
  - FERPA Family Education Rights and Privacy Act
  - COPPA Children's Online Privacy Protection Act

# **8 CONSENT OF ADULTS** Review the following definitions before answering the questions in this section. is the process of informing potential subjects about the research and asking them whether they want to participate. It usually (but not always) includes an opportunity **CONSENT** for subjects to ask questions. It does not necessarily include the signing of a consent form. This question is about the consent process. refers to how a subject's decision to participate in the research is documented. This is CONSENT DOCUMENTATION typically obtained by having the subject sign a consent form. is a document signed by subjects, by which they agree to participate in the research as **CONSENT FORM** described in the consent form and in the consent process. are specific information that is required to be provided to subjects. **ELEMENTS OF CONSENT** is the parent's active permission for the child to participate in the research. Parental PARENTAL PERMISSION permission is subject to the same requirements as consent, including written documentation of permission and required elements. is an alternative way of obtaining written documentation of consent that is most SHORT FORM CONSENT commonly used with individuals who are illiterate or whose language is one for which translated consent forms are not available. means there is IRB approval for not obtaining consent or for not including some of the elements of consent in the consent process. **WAIVER OF CONSENT** NOTE: If you plan to obtain identifiable information or identifiable biospecimens without consent, any waiver granted by the IRB does not override a subject's refusal to provide broad consent (for example, the Northwest Biotrust). WAIVER OF DOCUMENTATION means that there is IRB approval for not obtaining written documentation of consent. OF CONSENT **8.1 Groups** Identify the groups to which your answers in this section apply. Adult subjects Parents who are providing permission for their children to participate in research → If you selected **PARENTS**, the word "consent" below should also be interpreted as applying to parental permission and "subjects" should also be interpreted as applying to the parents. 8.2 The consent process. This series of questions is about whether you will obtain consent for all procedures except recruiting and screening and, if yes, how. The issue of consent for recruiting and screening activities is addressed in question 4.6. You do not need to repeat your answer to question 4.6.

a. Are there any procedures for which you will not obtain consent?

| No | Х |
|----|---|
| Ye | |

→ If yes, use the table below to identify the procedures for which you will not obtain consent. "All" is an acceptable answer for some studies.

Be sure to consider all research procedures and plans, including future contact, and sharing/banking of data and specimens for future work.

| Group¹ | Describe the procedures or data/specimen collection (if any) for which there will be NO consent process | Reason why you will not obtain<br>consent | Will<br>prov<br>subject<br>info abo<br>researc<br>they fi | vide<br>ts with<br>out the<br>th after |
|---|---|---|---|---|
| | | | YES | NO |

### Table footnotes

- 1. If your answer is the same for all groups you can collapse your answer across the groups and/or procedures.
  - **b.** <u>Describe the consent process</u>, if you will obtain consent for any or all procedures, for any or all groups. Address groups and procedures separately if the consent processes are different.

Be sure to include:

- The location/setting where consent will be obtained
- Who will obtain consent (refer to positions, roles, or titles, not names).
- Whether/how you will provide an opportunity for questions
- How you will provide an adequate opportunity for the subjects to consider all options

### Aim 1:

[redacted]

## Aims 2/3:

Local health departments that are interested in participating in the study will receive a written memorandum of understanding (MOU) that outlines the project, the research team's responsibilities, and the local health department's responsibilities. The local health department director and the staff person(s) who will participate in the study will sign the MOU. While not legally binding, a signed MOU provides a written record ensuring that (a) the director understands and supports staff member roles in the study and (b) the local health department staff member understands the scale of the training and *Connect to Wellness* goals. The MOU also documents everything UW will provide in terms of training, materials, and TA. We will consider a local health department enrolled in the study after it returns the signed MOU and one or more of their staff attends the first training session. Local health department staff will also be given an information sheet that outlines their responsibilities and contains additional elements of consent.

Worksite representatives will be provided with information about the brief satisfaction survey and asked if they would be willing to participate in the survey.

**c.** <u>Comprehension</u>. Describe how you will ensure or test the subjects' understanding of the information during the consent process.

We will ask participants if they have any questions and if they understand the purpose of the study/study procedures.

**d.** <u>Influence</u>. Does your research involve any subject groups that might find it difficult to say "no" to your research because of the setting or their relationship with you, even if you don't pressure them to participate?

Examples: Student participants being recruited into their teacher's research; patients being recruited into their healthcare provider's research, study team members who are participants; outpatients recruited from an outpatient surgery waiting room just prior to their surgery.



→ If yes, describe what you will do, for each of these subject groups, to reduce any effect of the setting or relationship on their decision.

Examples: a study coordinator will obtain consent instead of the subjects' physician; the researcher will not know which subjects agreed to participate; subjects will have two days to decide after hearing about the study.

**e.** Ongoing process. For research that involves multiple or continued interaction with subjects over time, describe the opportunities (if any) you will give subjects to ask questions or to change their minds about participating.

# Aim 1: [redacted]

Aims 2/3:

The local health department staff will be in regular monthly communication with members of the research team via technical assistance support and will be given opportunities to share their experiences with the study and decline to continue participation, if desired.

**8.3 Written documentation of consent.** Which of the statements below describe whether you will obtain documentation of consent? NOTE: This question does not apply to screening and recruiting procedures which have already been addressed in <u>question 4.6</u>.

Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent

**a.** Are you obtaining written documentation of consent for:

| None of your research procedures | → Use the table below to provide your justification then go to question<br>8.4. |
|---|---|
| All of your research procedures | → Do not complete the table; go to question 8.4. |
| Some of your research procedures | → Use the table below to identify the procedures for which you will<br>not obtain written documentation of consent from your adult<br>subjects. |

| Adult subject<br>group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO documentation of consent | Will<br>provide<br>with a v<br>stater<br>describi<br>resea<br>(optio | them written ment ing the arch |
|---|---|---|---|
| Aim 1: State chronic disease directors | We will conduct telephone interviews. | х | |
| Aim 1: Local health department directors | We will conduct telephone interviews. | х | |
| Aim 1: Local health department staff | We will conduct focus group discussions. | х | |
| Aims 2/3: Local<br>health department<br>staff | We will collect data from staff on their local health department's characteristics; satisfaction with training and technical assistance; implementation and intent to maintain <i>Connect to Wellness</i> ; and staff and worksite activities | х | |
| Aims 2/3: Worksite representatives | We will administer brief satisfaction surveys among a sample of worksites recruited by local health department staff. | x | |
| 8.4 Non-English-speaki fluency or literacy i x No Yes → If ye then to t | ing or -reading adult subjects. Will you enroll adult subjects who do not speak Engin English? es, describe the process you will use to ensure that the oral and written information during the consent process and throughout the study will be in a language reading and (for written materials such as consent forms or questionnaires) at an appending/comprehension level. | lish or who<br>on provided<br>ly underst | o lack<br>I to |
| a. <u>Interpretation</u> . Describe how you will provide interpretation and when. Also, describe the qualifications of the interpreter(s) – for example, background, experience, language proficiency in English and in the other language, certification, other credentials, familiarity with the research-related vocabulary in English and the target language. | | | |
| | <u>Translations</u> . Describe how you will obtain translations of all study materials (not just and how you will ensure that the translations meet the UW IRB's requirement that documents will be linguistically accurate, at an appropriate reading level for the papopulation, and culturally sensitive for the locale in which they will be used. | t translate | - |

- **8.5 Barriers to written documentation of consent**. There are many possible barriers to obtaining written documentation of consent. Consider, for example, individuals who are functionally illiterate; do not read English well; or have sensory or motor impairments that may impede the ability to read and sign a consent form.
  - **a.** Describe your plans (if any) for obtaining written documentation of consent from potential subjects who may have difficulty with the standard documentation process (that is, reading and signing a consent form). Skip this question if you are not obtaining written documentation of consent for any part of your research.

| you are not | obtaining written documentation of consent for any part of your research. |
|---|---|
| | f solutions: Translated consent forms; use of the Short Form consent process; reading the form to the person sign it; excluding individuals who cannot read and understand the consent form. |
| | 2/3, we will exclude local health departments whose local health department directors and staff cannot understand the MOU from the study. Given the study population, we do not anticipate that this will |
| "Blinding" subje | Il you deliberately withhold information or provide false information to any of the subjects? Note: ects to their study group/condition/arm is not considered to be deception. If yes, describe what information and why. Example: you may wish to deceive subjects about the purpose of the study. |
| | a. Will you debrief the subjects later? (Note: this is not required.) No Yes → If yes, describe how you will debrief the subjects. Upload any debriefing materials, including talking points or a script, to the Consent Form and Recruitment Materials SmartForm of Zipline. |
| 8.7 Cognitively impresearch? | paired adults, and other adults unable to consent. Do you plan to include such individuals in your |
| Examples: indivintoxicated. | viduals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are significantly |
| x No | → If no, go to <u>question 8.8</u> . |
| Yes | <ul> <li>→ If yes, answer the following questions.</li> <li>a. Rationale. Provide your rationale for including this population in your research.</li> </ul> |
| | b. <u>Capacity for consent / decision making capacity</u> . Describe the process you will use to determine whether a cognitively impaired individual is capable of consent decision making with respect to your research protocol and setting. |

| b.1. If you will have repeated interactions with the impaired subjects over a time period when cognitive capacity could increase or diminish, also describe how (if at all) you will reassess decision-making capacity and obtain consent during that time. |
|---|
| c. <u>Permission (surrogate consent)</u> . If you will include adults who cannot consent for themselves, describe your process for obtaining permission ("surrogate consent") from a legally authorized representative (LAR). |
| For research conducted in Washington State, see the <b>SOP: Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". |
| d. <u>Assent</u> . Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process you will use to obtain and document assent from the subjects. |
| e. <u>Dissent or resistance</u> . Describe how you will identify the subject's objection or resistance to participation (including non-verbal) during the research, and what you will do in response. |
| seems related restorials. Unlock to the Concept Forms and Doornitment Meterials ConcetForms of <b>7inling</b> all concept |

- **8.8 Consent-related materials.** Upload to the **Consent Forms and Recruitment Materials** SmartForm of **Zipline** all consent scripts/talking points, consent forms, debriefing statements, Information Statements, Short Form consent forms, parental permission forms, and any other consent-related materials you will use.
  - <u>Translations must be included</u>. However, you are strongly encouraged to wait to provide them until you know that the IRB will approve the English versions.
  - <u>Combination forms</u>: It may be appropriate to combine parental permission with consent, if parents are subjects as well as providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

## 9 PRIVACY AND CONFIDENTIALITY

**9.1 Privacy protections.** Describe the steps you will take, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection.

Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from medical
  records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the subject
  about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedures (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

Aim 1: [redacted]

For all aims, data will be stored on a secured server at UW. Files will not be identified by participant name.

**9.2 Identification of individuals in publications and presentations**. Do you plan to use potentially identifiable information about subjects in publications and presentations, or is it possible that individual identities could be inferred from what you plan to publish or present?



- **9.3** State mandatory reporting. Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:
  - Child abuse
  - · Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
  - Sexual assault
  - Serious physical assault
  - Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of your research team likely to learn of any of the above events or circumstances while conducting your research **AND** feel obligated to report it to state authorities?

| х | No | |
|---|---|---|
| | Yes | $\rightarrow$ If yes, the UW IRB expects you to inform subjects of this possibility in the consent form or during the |
| | | consent process, unless you provide a rationale for not doing so: |

(9.4) Retention of identifiers and data. Check the box below to indicate your assurance that you will not destroy any identifiers (or links between identifiers and data/specimens) and data that are part of your research records until after the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor; Food and Drug Administration) for your research. If you think it is important for your specific study to say something about destruction of identifiers (or links to identifiers) in your consent form, state something like "the link between your identifier and the research data will be destroyed after the records retention period required by state and/or federal law."

This question can be left blank for conversion applications (existing paper applications that are being "converted" into a Zipline application.)

See the "Research Data" sections of the following website for UW Records management for the Washington State research rectords retention schedules that apply in general to the UW (not involving UW Medicine data):

http://f2.washington.edu/fm/recmgt/gs/research?title=R

See the "Research Data and Records" information in Section 8 of this document for the retention schedules for UW Medicine Records: <a href="http://www.uwmedicine.org/about/Documents/UWM-Records-Retention-Schedule-v1.6.pdf">http://www.uwmedicine.org/about/Documents/UWM-Records-Retention-Schedule-v1.6.pdf</a>



**9.5** Certificates of Confidentiality. Are you planning to obtain a federal Certificate of Confidentiality for your research data? *NOTE: Answer "No" if your study is NIH funded, because all NIH-funded studies automatically have a Certificate.* 



- 9.6 Data and specimen security protections. Identify your data classifications and the security protections you will provide, referring to the <u>ZIPLINE GUIDANCE</u>: Data and Security Protections for the minimum requirements for each data classification level. You cannot answer this question without reading this document. Data security protections should not conflict with records retention requirements.
  - **a.** Which level of protections will you apply to your data and specimens? If you will use more than one level, describe which level will apply to which data and which specimens.

Level 1

**b.** Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. If there are any protections within the level listed in 9.6.a which you will *not* follow, list those here.

All project data will be stored on a secured server.
## **10 RISK / BENEFIT ASSESSMENT**

- **10.1** Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how you will manage or reduce the risks. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider possible physical, psychological, social, legal, and economic harms, including possible negative effects on financial standing, employability, insurability, educational advancement or reputation. For example, a breach of confidentiality might have these effects.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

The only risk associated with the study is a breach of confidentiality. This risk is small because security measures are in place to protect all data. Furthermore, the nature of the data gathered is not sensitive. No additional (e.g. physical) risks to subjects are anticipated. Datasets will use study IDs to further help protect participant confidentiality.

**10.2** Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.



No

→ If no go to question 10.3

Yes

→ If yes, answer the following questions:

a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks.

**b. Steps to minimize risk**. Describe the specific steps you will take to minimize the magnitude, probability, or duration of these risks.

Examples: inform the subjects about the risks and how to minimize them; require a pregnancy test before and during the study; require subjects to use contraception; advise subjects about banking of sperm and ova.

If you will require the use of contraception: describe the allowable methods and the time period when contraception must be used.

c. Pregnancy. Describe what you will do if a subject (or a subject's partner) becomes pregnant

For example; will you require the subject to immediately notify you, so that you can discontinue or modify the study procedures, discuss the risks, and/or provide referrals or counseling?

01/12/2018 Version 1.7

| 10.3 Unforeseeable risks | . Are there any research procedures that may have risks that are currently unforeseeable? |
|---|---|
| Example: using a drug | g that hasn't been used before in this subject population. |
| x No | |
| Yes $\rightarrow$ If y | yes, identify the procedures. |
| | e under regional or general anesthesiology. Will any research procedures occur while subjects- |
| patients are under g<br>(supplied for non-res | eneral or regional anesthesia, or during the 3 hours preceding general or regional anesthesia |
| x No | sedicit reasons). |
| | yes, check all the boxes that apply. |
| | Administration of any drug for research purposes |
| | Inserting an intra-venous (central or peripheral) or intra-arterial line for research purposes |
| | Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid for research purposes |
| | Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
| | Administration of a radio-isotope for research purposes** |
| | Implantation of an experimental device |
| | Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |
| | If you checked any of the boxes: You must provide the name and institutional affiliation of a physician anesthesiologist who is a member of your research team or who will serve as a safety consultant about the interactions between your research procedures and the general or regional anesthesia of the subject-patients. If your procedures will be performed at a UW Medicine facility or affiliate, the anesthesiologist must be a UW faculty member. |
| | ** If you checked the box about radio-isotopes: you are responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval. |
| NIH). If required for | <b>nitoring</b> . A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined by your research, upload your DSMP to the <b>Supporting Documents</b> SmartForm in <b>Zipline</b> . If it is er document you are uploading (for example, a Study Protocol, use the text box below to name the DSMP. |
| N/A | |

| N/A | |
|---|---|
| withdrawn from t<br>participant, regar | rticipants. If applicable, describe the anticipated circumstances under which participants will be the research without their consent. Also, describe any procedures for orderly withdrawal of a dless of the reason, including whether it will involve partial withdrawal from procedures and any continued data collection or long-term follow-up. |
| N/A | |
| / | t benefits to participants. If there are any direct research-related benefits that some or all individual kely to experience from taking part in the research, describe them below: |
| | refits to society or others, and do not include subject payment (if any). Examples: medical benefits such as subjects receive the results); psychological resources made available to participants; training or education |
| Aim 1:<br>[redacted] | |
| | nefit to local health departments is increased capacity to do worksite wellness activities. Worksites<br>kers will potentially benefit from this research by creating healthier environments for their workers. |
| 9 Individual subject | s findings. |
| | at your research will unintentionally discover a previously unknown condition such as a disease, |
| Suicidal III | entions, or genetic predisposition? |
| x No | entions, or genetic predisposition? |
| x No<br>Yes<br>b. Do you plar | → If yes, explain whether and how you would share the information with the subject. |
| x No<br>Yes b. Do you plar<br>genetic tes | entions, or genetic predisposition? → If yes, explain whether and how you would share the information with the subject. It to share the individual results of any of your study procedures or findings with the subjects — such as |
| x No<br>Yes b. Do you plar<br>genetic tes | entions, or genetic predisposition? → If yes, explain whether and how you would share the information with the subject. It to share the individual results of any of your study procedures or findings with the subjects — such as tresults, laboratory tests, etc.? |
| b. Do you plar genetic test You should to Yes | <ul> <li>→ If yes, explain whether and how you would share the information with the subject.</li> <li>It is share the individual results of any of your study procedures or findings with the subjects – such as a results, laboratory tests, etc.?</li> <li>If yes, complete and upload the SUPPLEMENT: Participant Results Sharing to the Supporting</li> </ul> |
| b. Do you plar genetic test You should to X No Yes 10 Commercial pro x No | <ul> <li>→ If yes, explain whether and how you would share the information with the subject.</li> <li>It is share the individual results of any of your study procedures or findings with the subjects – such as tresults, laboratory tests, etc.?</li> <li>If yes, complete and upload the SUPPLEMENT: Participant Results Sharing to the Supporting Documents SmartForm of Zipline</li> </ul> |

## 11 ECONOMIC BURDEN TO PARTICIPANTS

**11.1 Financial responsibility for research-related injuries.** Answer this question only if the lead researcher is <u>not</u> a UW student, staff member, or faculty member whose primary paid appointment is at the UW.

Describe who will be financially responsible for research-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which participants may obtain treatment/compensation.

N/A

11.2 Costs to subjects. Describe any research-related costs for which subjects and/or their health insurance may be responsible (examples might include: CT scan required for research eligibility screening; co-pays; surgical costs when a subject is randomized to a specific procedure; cost of a device; travel and parking expenses that will not be reimbursed).

Aims 2/3:

Local health department staff will be responsible for costs related to travel (e.g. going to meet with a worksite) and printing materials for worksites (e.g. *Connect to Wellness* intervention toolkits).

11.3 Reimbursement for costs. Describe any costs to subjects that will be reimbursed (such as travel expenses).

Aims 2/3:

Local health department staff will not be reimbursed for any costs.

### **12 RESOURCES**

- **12.1** Faculty Advisor. (For researchers who are students, fellows, or post-docs.) Provide the following information about your faculty advisor.
  - Advisor's name
  - Your relationship with your advisor (for example: graduate advisor; course instructor)
  - Your plans for communication/consultation with your advisor about progress, problems, and changes.

N/A

**12.2 Study team communication**. Describe how you will ensure that each study team member is adequately trained and informed about the research procedures and requirements (including any changes) as well as their research-related duties and functions.

There is no study team.

All of the investigators on the study team have been trained on IRB, and we will ensure that all study staff have up to date training prior to contacting any participants. The study team will meet at least every other week throughout the project. Study materials will be stored on a shared drive to ensure that all members have ready access to the latest protocols, instruments, and other project-related materials.

# 13 OTHER APPROVALS, PERMISSIONS, and REGULATORY ISSUES

**13.1 Other regulatory approvals**. Identify any other regulatory approvals that are required for this research, by checking applicable boxes

Do not attach the approvals unless requested by the IRB.

| | Approval | Research for which this is required |
|---|---|---|
| Radiation | ı Safety | Procedures involving the use of radioactive materials or an ionizing radiatio producing machine radiation, if they are conducted for research rather than clinical purposes. Approvals need to be attached to the Supporting Documents page in <i>Zipline</i> . |
| Institution | nal Biosafety | Procedures involving the transfer/administration of recombinant DNA, DNA/RNA derived from recombinant DNA, or synthetic DNA. |
| RDRC | | Procedures involving a radioactive drug or biological product that is not approved by the FDA for the research purpose and that is being used witho an IND, for basic science research (not to determine safety and effectiveness or for immediate therapeutic or diagnostic purposes). |
| ESCRO | | Procedures involving the use of some types of human embryonic stem cells |
| Do not attach | n the approvals and permissic | ng agency, employee union, UW Medicine clinical unit. ons unless requested by the IRB. |
| Do not attach | n the approvals and permissio | |
| N/A<br>Financial Cor | | member of the team have a Financial Conflict of Interest (FCOI) in this |

### **Study Identification**

Unique protocol identification number: STUDY00004627

Brief Title: Training LHD's to disseminate evidence-based interventions to small work sites

Official Training Local Health Departments to Disseminate Evidence-Based Interventions to Small and

Title: Low-Wage Worksites

Secondary 2R01CA160217 [U.S. NIH Grant/Contract Award Number]

IDs: NCI-2021-02876 [Registry ID: CTRP (Clinical Trial Reporting Program)]

RG1121453 [Fred Hutch/University of Washington Cancer Consortium]

### Document date: June 10, 2020

The protocol reviewed by the University of Washington Institutional Review Board appears below. Information about an additional study (Aim 1 activities in the protocol) outside of the randomized trial and information that describes individuals' names or intellectual property has been redacted.





## **INSTRUCTIONS**

- <u>If you are requesting a determination</u> about whether your activity is human subjects research or qualifies for exempt status, you may skip all questions except those marked with a . For example 1.1 must be answered.
- Answer all questions. If a question is not applicable to your research or if you believe you have already answered a question elsewhere in the application, state "NA" (and if applicable, refer to the question where you provided the information). If you do not answer a question, the IRB does not know whether the question was overlooked or whether it is not applicable. This may result in unnecessary "back and forth" for clarification. Use non-technical language as much as possible.
- To check a box, place an "X" in the box. To fill in a text box, make sure your cursor is within the gray text box bar before typing or pasting text.
- The word "you" refers to the researcher and all members of the research team, unless otherwise specified.
- For collaborative research, describe only the information that is relevant to you unless you are requesting that the UW IRB provide the review and oversight for your collaborators as well.
- You may reference other documents (such as a grant application) if they provide the requested information in non-technical language. Be sure to provide the document name, page(s), and specific sections, and upload it to *Zipline*. Also, describe any changes that may have occurred since the document was written (for example, changes that you've made during or after the grant review process). In some cases, you may need to provide additional details in the answer space as well as referencing a document.

| INDEX | | |
|---|---|---|
| 1 Overview | 6 Children (Minors) and Parental Permission | 10 Risk / Benefit Assessment |
| 2 Participants | 7 Assent of Children (Minors) | 11 Economic Burden to Participants |
| 3 Non-UW Research Setting | 8 Consent of Adults | 12 Resources |
| 4 Recruiting and Screening Participants | 9 Privacy and Confidentiality | 13 Other Approvals, Permissions, and Regulatory Issues |

## 1 OVERVIEW

**Study Title:** 

Disseminating Connect to Wellness Via Local Health Departments

1.1)Home institution. Identify the institution through which the lead researcher listed on the IRB application will conduct the research. Provide any helpful explanatory information.

In general, the home institution is the institution (1) that provides the researcher's paycheck and that considers him/her to be a paid employee, or (2) at which the researcher is a matriculated student. Scholars, faculty, fellows, and students who are visiting the UW and who are the lead researcher: identify your home institution and describe the purpose and duration of your UW visit, as well as the UW department/center with which you are affiliated while at the UW.

Note that many UW clinical faculty members are paid employees of non-UW institutions.

The UW IRB provides IRB review and oversight for only those researchers who meet the criteria described in the POLICY: Use of the UW IRB.

University of Washington

1.2)Consultation history. Have you consulted with anyone at HSD about this study?

It is not necessary to obtain advance consultation. If you have: answering this question will help ensure that the IRB is aware of and considers the advice and guidance you were provided.



No

→ If yes, briefly describe the consultation: approximate date, with whom, and method (e.g. by email, phone call, in-person meeting).

We discussed this study with [redacted] via e-mail on 3/30/18 and 4/2/18, and via telephone on 8/21/2018. We also consulted with [redacted] via phone and e-mail in July/August 2019.

1.3) Similar and/or related studies. Are there any related IRB applications that provide context for the proposed activities?

Examples of studies for which there is likely to be a related IRB application: Using samples or data collected by another study; recruiting subjects from a registry established by a colleague's research activity; conducting Phase 2 of a multi-part project, or conducting a continuation of another study; serving as the data coordinating center for a multi-site study that includes a UW site.

Providing this information (if relevant) may significantly improve the efficiency and consistency of the IRB's review.



→ If yes, briefly describe the other studies or applications and how they relate to the proposed activities. If the other applications were reviewed by the UW IRB, please also provide: the UW IRB number, the study title, and the lead researcher's name.

The current IRB application is for a National Cancer Institute funded competing renewal of our HealthLinks R01 (grant number R01CA160217). The former proposal was to test the effectiveness of the HealthLinks intervention for small worksites. The IRB number was 45447EJ, study title: HealthLinks Trial: Increasing Implementation of Evidence-Based Interventions at Low-Wage Worksites, and the lead researcher was Margaret (Peggy) Hannon.

Please note that we changed the name of the intervention for the current project and IRB proposal. We learned that the name HealthLinks was trademarked by another group, and changed the name to Connect to Wellness. However, the intervention is the same.

Finally, the current IRB application is related to application number 00004627, which we submitted in April 2018 as part of our Just In Time package to NCI and modified for our initial study in November 2018 and August 2019.

1.4) Externally-imposed urgency or time deadlines. Are there any externally-imposed deadlines or urgency that affect your proposed activity?

HSD recognizes that everyone would like their IRB applications to be reviewed as quickly as possible. To ensure fairness, it is HSD policy to review applications in the order in which they are received. However, HSD will assign a higher priority to research with externally-imposed urgency that is beyond the control of the researcher. Researchers are encouraged to communicate as soon as possible with their HSD staff contact person when there is an urgent situation (in other words, before submitting the IRB application). Examples: a researcher plans to test an experimental vaccine that has just been developed for a newly emerging epidemic; a researcher has an unexpected opportunity to collect data from students when the end of the school year is only four weeks away.

HSD may ask for documentation of the externally-imposed urgency. A higher priority should not be requested to compensate for a researcher's failure to prepare an IRB application in a timely manner. Note that IRB review requires a certain minimum amount of time; without sufficient time, the IRB may not be able to review and approve an application by a deadline.



No

→ If yes, briefly describe the urgency or deadline as well as the reason for it.

1.5)Objectives Using lay language, describe the purpose, specific aims, or objectives that will be met by this specific project. If hypotheses are being tested, describe them. You will be asked to describe the specific procedures in a later section.

If your application involves the use of a HUD "humanitarian" device: describe whether the use is for "on-label" clinical patient care, "off-label" clinical patient care, and/or research (collecting safety and/or effectiveness data).

The primary goals of this study are to (a) scale up Connect to Wellness by training staff in local health departments across the United States to deliver Connect to Wellness to small worksites in their communities, and (b) conduct a trial comparing the effectiveness and costs of two different implementation strategies.

It has been previously proven that Connect to Wellness is effective. Our objective now is to determine the best way to implement it. Although the local health departments will be involved in collecting identifiable data, they are not engaged in the research because we are not testing the efficacy of Connect to Wellness.

Study goals will be achieved through three aims:

Aim 1: Conduct formative research (interviews and focus groups) with state and local health departments Aim 2: Test two different implementation strategies with local health departments: 1) standard Connect to Wellness training and technical assistance and 2) standard Connect to Wellness training plus enhanced technical assistance Aim 3: Measure the costs of each implementation strategy

**1.6) Study design**. Provide a one-sentence description of the general study design and/or type of methodology.

Your answer will help HSD in assigning applications to reviewers and in managing workload. Examples: a longitudinal observational study; a double-blind, placebo-controlled randomized study; ethnographic interviews; web scraping from a convenience sample of blogs; medical record review; coordinating center for a multi-site study.

Aim 1 activities are qualitative. We will conduct semi-structured interviews and focus groups with participants via online and telephone methods.

Aim 2 is a hybrid type III randomized controlled trial comparing two different Connect to Wellness implementation strategies. We will randomize 40 local health departments to receive either a 1) standard training and technical assistance or 2) standard training plus enhanced technical assistance.

Aim 3 will measure the costs associated with each implementation strategy via process measures (e.g. tracking worksheets) and conduct a cost analysis based on this data.

(1.7)Intent. Check all the descriptors that apply to your activity. You must place an "X" in at least one box.

This question is essential for ensuring that your application is correctly reviewed. Please read each option carefully.

| Descriptor |
|---|
| 1. Class project or other activity whose purpose is to provide an educational experience for the researcher (for example, to learn about the process or methods of doing research). |
| 2. Part of an institution, organization, or program's own internal operational monitoring. |
| 3. Improve the quality of service provided by a specific institution, organization, or program. |
| 4. Designed to expand the knowledge base of a scientific discipline or other scholarly field of study, and produce results that: |
| <ul> <li>Are expected to be applicable to a larger population beyond the site of data collection or the specific<br/>subjects studied, or</li> </ul> |
| <ul> <li>Are intended to be used to develop, test, or support theories, principles, and statements of relationships,<br/>or to inform policy beyond the study.</li> </ul> |
| 5. Focus directly on the specific individuals about whom the information or biospecimens are collected through oral history, journalism, biography, or historical scholarship activities, to provide an accurate and evidence-based portrayal of the individuals. |
| 6. A quality improvement or program improvement activity conducted to improve the implementation (delivery or quality) of an accepted practice, or to collect data about the implementation of the practice for clinical, practical, or administrative purposes. This does not include the evaluation of the efficacy of different accepted practices, or a comparison of their efficacy. |
| 7. Public health surveillance activities conducted, requested, or authorized by a public health authority for the sole purpose of identifying or investigating potential public health signals or timely awareness and priority setting during a situation that threatens public health. |
| 8. Preliminary, exploratory, or research development activities (such as pilot and feasibility studies, or reliability/validation testing of a questionnaire) |
| 9. Expanded access use of a drug or device not yet approved for this purpose |
| 10. Use of a Humanitarian Use Device |
| 11. Other. Explain: |

- **1.8 Background, experience, and preliminary work**. Answer this question <u>only</u> if your proposed activity has one or more of the following characteristics. The purpose of this question is to provide the IRB with information that is relevant to its risk/benefit analysis.
  - Involves more than minimal risk (physical or non-physical)
  - Is a clinical trial, or
  - Involves having the subjects use a drug, biological, botanical, nutritional supplement, or medical device.

"Minimal risk" means that the probability and magnitude of harm or discomfort anticipated in the research are not greater than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests.

**a.** <u>Background</u>. Provide the rationale and the scientific or scholarly background for your proposed activity, based on existing literature (or clinical knowledge). Describe the gaps in current knowledge that your project is intended to address.

This should be a plain language description. Do not provide scholarly citations. Limit your answer to less than one page, or refer to an attached document with background information that is no more than three pages long.

Cancer and other chronic diseases are the leading causes of death in the United States. Several preventable risk behaviors, including physical inactivity, unhealthy eating, missed cancer screenings, and tobacco use increase disease risk. Evidence-based interventions significantly reduce each of these risk behaviors. Most adults in the United States are employed, and worksites can implement evidence-based interventions to support worker health.

However, small worksites (businesses with less than 250 employees) infrequently implement these interventions and face budget, capacity, and partnership challenges in doing so. To assist these worksites, we previously partnered with the American Cancer Society to create and test *Connect to Wellness*, a program to disseminate evidence-based interventions and provide implementation support. The findings from this work show that *Connect to Wellness* is effective, but wider dissemination of this program has yet to occur.

Local health departments cover most communities, and most local health department goals include preventing chronic disease. Previous studies of local health department activities and investments show positive associations between their efforts and health outcomes in communities. Given this information, these departments have the potential to assist with the dissemination of *Connect to Wellness* nationwide. While local health departments are a vital part of community-based chronic disease practice, they are underrepresented in implementation research.

**b.** Experience and preliminary work. Briefly describe experience or preliminary work or data (if any) that you or your team have that supports the feasibility and/or safety of this study.

It is not necessary to summarize all discussion that has led to the development of the study protocol. The IRB is interested only in short summaries about experiences or preliminary work that suggest the study is feasible and that risks are reasonable relative to the benefits. Examples: You have already conducted a Phase 1 study of an experimental drug which supports the Phase 2 study you are now proposing to do; you have already done a small pilot study showing that the reading skills intervention you plan to use is feasible in an after-school program with classroom aides; you have experience with the type of surgery that is required to implant the study device; you have a study coordinator who is experienced in working with subjects who have significant cognitive impairment.

We previously tested the *Connect to Wellness* intervention in a pilot study and randomized controlled trial. In 2012, we trained a health educator in a rural local health department to deliver *Connect to Wellness*. Training included in-person meetings and observations. To make training and technical assistance more sustainable, we

developed and pilot-tested a distance-training model with success in several local health departments in Washington State.

**1.9 Supplements**. Check all boxes that apply, to identify Supplements you should complete and upload to the **Supporting Documents** SmartForm in *Zipline*.

This section is here instead of at the end of the form to reduce the risk of duplicating information in this IRB Protocol form that you will need to provide in these Supplements.

| Check all<br>That Apply | Type of Research | Supplement Name |
|---|---|---|
| | <b>Department of Defense</b> The research involves Department of Defense funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Defense |
| | <b>Department of Energy</b> The research involves Department of Energy funding, facilities, data, or personnel. | ZIPLINE SUPPLEMENT: Department of Energy |
| | <b>Drug, biologic, botanical, supplement</b> Procedures involve the use of <u>any</u> drug, biologic, botanical or supplement, even if the item is not the focus of your research | ZIPLINE SUPPLEMENT: Drugs |
| | Emergency exception to informed consent Research that requires this special consent waiver for research involving more than minimal risk | ZIPLINE SUPPLEMENT: Exception from Informed Consent for Emergency Research (EFIC) |
| | Genomic data sharing Genomic data are being collected and will be deposited in an external database (such as the NIH dbGaP database) for sharing with other researchers, and you are asking the UW to provide the required certification or to ensure that the consent forms can be certified | ZIPLINE SUPPLEMENT: Genomic Data Sharing |
| | <b>Medical device</b> Procedures involve the use of <u>any</u> medical device, even if the device is not the focus of your research, except when the device is FDA-approved and is being used through a clinical facility in the manner for which it is approved | ZIPLINE SUPPLEMENT: Devices |
| | Multi-site study (You are asking the UW IRB to review one or more sites in a multi-site study.) | ZIPLINE SUPPLEMENT: Participating Site in Multi- Site Research |
| | Participant results sharing Individual research results will be shared with subjects. | ZIPLINE SUPPLEMENT:<br>Participant Results<br>Sharing |
| х | None of the above | |

## **2 PARTICIPANTS**

| health status, and any other relevant characteristics. |
|---|
| Aim 1: [redacted] Aims 2/3: The first group of participants will be <u>local health department staff</u> , coming from 40 local health departments across the U.S., who will be trained to recruit and deliver Connect to Wellness to small worksites in their communities. The second group of participants will be <u>representatives from these worksites</u> , who will provide feedback about their experiences with Connect to Wellness via a brief satisfaction survey. To conduct the cost analysis for Aim 3, we will use data collected by members of the research team and by local health department staff. |
| 2.2) nclusion and exclusion criteria. |
| <b>a. Inclusion criteria.</b> Describe the specific criteria you will use to decide who will be included in your study from among interested or potential subjects. Define any technical terms in lay language. |
| Aim 1: [redacted] Aims 2/3: Local health departments in the 50 states and District of Columbia will be eligible to participate in the randomized controlled trial. Additional eligibility criteria include willingness to support one or more staff members to participate in <i>Connect to Wellness</i> training and the project for two years, and to have these staff recruit 15 or more worksites for <i>Connect to Wellness</i> over 24 months. We will recommend to local health department staff that they focus on recruiting worksites with 20-200 employees (i.e. worksites with fewer resources for workplace health promotion, and for which the strongest evidence for the effectiveness of <i>Connect to Wellness</i> is present). The worksite representatives will need to be able to speak and read English, and be knowledgeable about health and wellness at the worksite (e.g. HR manager). We expect that representatives will be at least 18 years of age or older. |
| b. Exclusion criteria. Describe the specific criteria you will use to decide who will be excluded from your study from subjects who meet the inclusion criteria listed above. Define any technical terms in lay language. |
| Aim 1: [redacted] Aims 2/3: Local health departments who are not able to support staff to participate in <i>Connect to Wellness</i> will be excluded from the study. |
| <b>2.3 Prisoners</b> . IRB approval is required in order to include prisoners in research, even when prisoners are not an intended target population. |
| a. Will you recruit or obtain data from individuals that you know to be prisoners? |
| For records reviews: if the records do not indicate prisoner status and prisoners are not a target population, select "No". See the <u>WORKSHEET: Prisoners</u> for the definition of "prisoner". |
| x No Yes → If yes, answer the following questions (i – iv). |
| i. Describe the type of prisoners, and which prisons/jails: |

| living conditions, medical care, qual | h is whether the effect of participation on prisoners' general ity of food, amenities, and opportunity for earnings in prison ifficult for prisoners to adequately consider the research risks. |
|---|---|
| | ure that (a) your recruitment and subject selection procedures nd (b) prison authorities or other prisoners will not be able to ular prisoners from participating. |
| Washington State: check the box be or facilitate the use of a prisoner's p | rs in federal facilities or in state/local facilities outside of<br>slow to provide your assurance that you will (a) not encourage<br>participation in the research to influence parole decisions, and<br>dvance (for example, in a consent form) that participation in<br>his or her parole. |
| Confirmed | |
| <b>b.</b> Is your research likely to have subjects who become | prisoners while participating in your study? |
| For example, a longitudinal study of youth with drug pr point during the study. | oblems is likely to have subjects who will be prisoners at some |
| procedures and/or data collection w | r while participating in your study, will you continue the study hile the subject is a prisoner? ocedures and/or data collection you will continue with prisoner |
| 2.4 Protected populations. IRB approval is required for the usany of these populations that you will purposefully include population is an inclusion criterion for your study.) | se of the subject populations listed here. Check the boxes for de in your research. (In other words, being a part of the |
| The WORKSHEETS describe the criteria for approval but do i | |
| Population | Worksheet |
| Fetuses in utero | WORKSHEET: Pregnant Women |
| Neonates of uncertain viability | WORKSHEET: Neonates |
| Non-viable neonates | WORKSHEET: Neonates |
| Pregnant women | WORKSHEET: Pregnant Women |

| | non U.S. indigenous populations. Will you actively recruit from Native American or non-U.S. ons through a tribe, tribe-focused organization, or similar community-based organization? |
|---|---|
| | e defined in international or national legislation as having a set of specific rights based on their historica<br>Pritory and their cultural or historical distinctiveness from other populations that are often politically |
| Examples: a reservat | ion school or health clinic; recruiting during a tribal community gathering |
| x No | |
| | , name the tribe, tribal-focused organization, or similar community based organization. The UW IF<br>cts that you will obtain tribal/indigenous approval before beginning your research. |
| САВС | and that you thin obtain thou, margemous approval service segmining your research |
| 'hind vantu avlaiasta | Will you called write identifiable information about ather individuals from your subjects? |
| | Will you collect private identifiable information about other individuals from your subjects? nclude: collecting medical history information or contact information about family members, |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest | |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest | nclude: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest readily identify the grown of the composition of the | nclude: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you and parents, then you are not collecting private identifiable information about the grandparents. es, these individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you andparents, then you are not collecting private identifiable information about the grandparents. These individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of the research team to read subjects several quest readily identify the grown as the readily identified in the readily identified in th | include: collecting medical history information or contact information about family members, any direct or indirect identifier that, alone or in combination, would allow you or another member of you lily identify the person. For example, suppose that you are studying immigration history. If you ask your ions about their grandparents but you do not obtain names or other information that would allow you and parents, then you are not collecting private identifiable information about the grandparents. es, these individuals are considered human subjects in your study. Describe them and what data will collect about them. |
| Common examples in friends, co-workers. "Identifiable" means of research team to reach subjects several quest readily identify the grown of the composition of the | nclude: collecting medical history information or contact information any direct or indirect identifier that, alone or in combination, would alloudily identify the person. For example, suppose that you are studying imnions about their grandparents but you do not obtain names or other information and parents, then you are not collecting private identifiable information es, these individuals are considered human subjects in your study. D |

# **2.7 Number of subjects.** Can you predict or describe the maximum number of subjects (or subject units) you need to complete your study, for each subject group?

<u>Subject units</u> mean units within a group. For most research studies, a group will consist of individuals. However, the unit of interest in some research is not the individual. Examples:

- Dyads such as caregiver-and-Alzheimer's patient, or parent and child
- Families
- Other units, such as student-parent-teacher

<u>Subject group</u> means categories of subjects that are meaningful for your research. Some research has only one subject group – for example, all UW students taking Introductory Psychology. Some common ways in which subjects are grouped include:

- By intervention for example, an intervention group and a control group.
- By subject population or setting for example, urban versus rural families
- By age for example, children who are 6, 10, or 14 years old.

The IRB reviews the number of subjects you plan to study in the context of risks and benefits. You may submit a Modification to increase this number at any time after you receive IRB approval. If the IRB determines that your research involves no more than minimal risk: you may exceed the approved number and it will not be considered non-compliance. If your research involves more than minimal risk: exceeding the approved number will be considered non-compliance.



→ If no, provide your rationale in the box below. Also, provide any information you can about the scope/size of the research. You do not need to complete the table.

Example: you may not be able to predict the number of subjects who will complete an online survey advertised through Craigslist, but you can state that you will post your survey for two weeks and the number who respond is the number who will be in your study.



→ If yes, for each subject group, use the table below to provide your estimate of the maximum desired number of individuals (or other subject unit, such as families) who will complete the research.

| research<br>*For clinical trials: provide numbers for your site and for<br>the study-wide total number |
|---|
| 25 |
| 40 |
| 80 |
| 40-80 |
| 600 |
| 2 4 4 |

# **3 NON-UW RESEARCH SETTING**

## Complete this section only if your research will take place outside of UW and Harborview

| Intext. Culturally-appropriate procedures and an understanding of local context are an important part of ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. Ses: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male their; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. Secific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: Secific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: Secific laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. Secific laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. Seally authorized representative — laws about who can serve as a legally authorized representative (and we spriority when more than one person is available) vary across states and countries. |
|---|
| ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. es: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male her; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. eral site maintains an international list of human research standards and requirements: www.hhs.gov/ohrp/international/index.html ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. eally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ing subjects. Describe any site-specific cultural issues, customs, beliefs, or values that may affect your research it is conducted. es: It would be culturally inappropriate in some international settings for a woman to be directly contacted by a male her; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. eral site maintains an international list of human research standards and requirements: www.hhs.gov/ohrp/international/index.html ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. eally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ther; instead, the researcher may need to ask a male family member for permission before the woman can be ched. It may be appropriate to obtain permission from community leaders prior to obtaining consent from individual rs of a group. The property of a group. The property of the maintains an international list of human research standards and requirements: The property of the provide consent vary ross states, and across countries. The property of the property of the property of the property of the property of the provide consent vary ross states, and across countries. The property of the property of the property of the property of the provide consent vary ross states, and across countries. The property of the property of the property of the provide consent vary ross states, and across countries. The property of the property of the property of the provide consent vary ross states, and across countries. |
| ecific laws. Describe any local laws that may affect your research (especially the research design and consent ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary ross states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and we |
| ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary oss states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and w |
| ures). The most common examples are laws about: ecimens – for example, some countries will not allow biospecimens to be taken out of the country. e of consent – laws about when an individual is considered old enough to be able to provide consent vary oss states, and across countries. gally authorized representative – laws about who can serve as a legally authorized representative (and w |
| e of healthcare records – many states (including Washington State) have laws that are similar to the deral HIPAA law but that have additional requirements. |
| ecific administrative or ethical requirements. Describe local administrative or ethical requirements that affect search. |
| e: A school district may require you to obtain permission from the head district office as well as school principals befo<br>ching teachers or students; a factory in China may allow you to interview factory workers but not allow you to pay |
| e :: |

**4.1** Recruiting and Screening. Describe how you will identify, recruit, and screen subjects. Include information about: how, when, where, and in what setting. Identify who (by position or role, not name) will approach and recruit subjects, and who will screen them for eligibility.

# Aim 1: [redacted]

#### Aims 2/3:

To recruit local health departments for the trial, The National Association for Chronic Disease Directors will include us on the agenda for a webinar or in-person meeting of the state chronic disease directors. To ensure outreach to the entire group, follow-up email communication will go to the state-level voting members. At the meeting, we will present *Connect to Wellness* and its evidence-base and describe the proposed trial. We will request that state chronic disease directors share this information with their local health departments, and will offer to follow-up individually if they have questions or concerns. We will work the state chronic disease directors who believe one or more local health departments in their state would be interested in the study to identify the best ways to recruit these local health departments. The state chronic disease director may make a referral to the local health department, linking their director or appropriate staff to the research team, or s/he may prefer to send out recruitment materials to local health department directors directly. If this approach does not yield 40 local health departments, we may use one or more of the following strategies to reach local health department directors directly: The director of the UW's Public Health Training Center, the Northwest Center for Public Health Practice, is a co-investigator for this study and is able to refer us to local health department directors in the multi-state region served by her Center. We may also advertise the study through the National Association of City and County Health Officials and/or through the Association of State and Territorial Health Officials (email blast or newsletter).

Recruitment materials will direct local health department directors or staff to contact a member of our research team via telephone for more information. Local health departments who contact us will be given more information about the study so that they understand the project purpose and duration, requirements of staff time, recruitment expectations, and data requirements. This conversation will serve as part of the screening process, whereby local health departments who cannot dedicate the staff and time to this project will not be invited to participate in the trial.

To recruit worksite representatives for the brief satisfaction survey, we will generate a random sample of five worksites per local health department (e.g. via a random numbers table) and contact representatives by e-mail or telephone to schedule a time to complete the brief satisfaction survey.

### 4.2 Recruitment materials.

a. What materials (if any) will you use to recruit and screen subjects?

Examples: talking points for phone or in-person conversations; video or audio presentations; websites; social media messages; written materials such as letters, flyers for posting, brochures, or printed advertisements; questionnaires filled out by potential subjects.

#### Aim 1:

[redacted]

### Aims 2/3:

We will have presentation materials (e.g. PowerPoint, talking points, and notes) to do initial outreach with state chronic disease directors. We will use written materials and a telephone script to talk to interested local health departments about the study. The content of the written materials will also reside on a website about *Connect to Wellness* for the recruitment phase.

b. Upload descriptions of each type of material (or the materials themselves) to the Consent Forms and Recruitment Materials SmartForm of **Zipline**. If you will send letters to the subjects, the letter should include a statement about how you obtained the subject's name, contact information, and any other subject-specific information (such as a health condition) that is mentioned in the letter.

HSD encourages researchers to consider uploading descriptions of most recruitment and screening materials instead of the materials themselves. The goal is to provide the researchers with the flexibility to change some information on the materials without submitting a Modification for IRB approval of the changes. Examples:

- You could provide a list of talking points that will be used for phone or in-person conversations instead of a script.
- For the description of a flyer, you might include the information that it will provide the study phone number and the name of a study contact person (without providing the actual phone number or name). In doing so, you would not need to submit a Modification if/when the study phone number or contact person changes. Also, instead of listing the inclusion/exclusion criteria, you might state that the flyer will list one or a few of the major inclusion/exclusion
- For the description of a video or a website, you might include a description of the possible visual elements and a list of the content (e.g., study phone number; study contact person; top three inclusion/exclusion criteria; payment of \$50; study name; UW researcher).
- 4.3 Relationship with participant population. Do any members of the study team have an existing relationship with the study population(s)?

Examples: a study team member may have a dual role with the study population (for example, being their clinical care provider, teacher, laboratory directory or tribal leader in addition to recruiting them for his/her research).



No

→ If yes, describe the nature of the relationship.

[redacted] at the National Association of Chronic Disease Directors (a co-investigator on the grant) consults with state-level public health leaders to improve their organization's practices. [redacted] (also a co-investigator on this grant) works for the Northwest Center for Public Health Practice, which provides training to local health departments. Neither manage or have direct oversight of individuals working in these settings.

- **4.4 Payment to participants**. Describe any payment you will provide, including:
  - The total amount/value
  - Whether payment will be "pro-rated" so that participants who are unable to complete the research may still receive some part of the payment

The IRB expects the consent process or study information provided to the subjects to include information about the number and amount of payments, and especially the time when subjects can expect to receive payment. One of the most frequent complaints received by HSD is from subjects who expected to receive cash or a check on the day that they completed a study and who were angry or disappointed when payment took 6-8 weeks to reach them.

Do not include a description of any expenses that will be reimbursed.

| N. | / A |
|----|-----|
| N | / A |

| | stude | nts; a | tary compensation. Describe any non-monetary compensation you will provide. Example: extra credit for toy for a child. If you will be offering class credit to students, you must provide (and describe) an alternate students to earn the extra credit without participating in your research. |
|---|---|---|---|
| | N/A | | |
| 4.6 | Will y | ou ac | cess or obtain data or specimens for recruiting and screening procedures prior to enrollment? |
| | | ionnai | ames and contact information; the information gathered from records that were screened; results of screening res or screening blood tests; Protected Health Information (PHI) from screening medical records to identify possible |
| | | No | → If no, skip the rest of this section; go to question 5.1. |
| | х | Yes | → If yes, describe any data and/or specimens (including PHI) you will access or obtain for recruiting and screening and whether you will retain it as part of the study data. |
| | | | Aim 1:<br>[redacted] |
| | | | Aims 2/3: We may obtain the names and contact information for individuals within the local health departments from the state chronic disease directors, should the director provide a referral for us. |
| 4.7 | | | r recruiting and screening. Will you obtain consent for any of the recruiting and screening procedures? Consent of Adults asks about consent for the main study procedures). |
| | | | ncludes: consent from individuals for their own participation; parental permission; assent from children; consent<br>Ily authorized representative for adult individuals who are unable to provide consent. |
| | •<br>•<br>• | Foi<br>fro<br>Foi<br>Foi | r a study in which names and contact information will be obtained from a registry: the registry should have consent m the registry participants to release their names and contact information to researchers. r a study in which possible subjects are identified by screening records: there will be no consent process. r a study in which individuals respond to an announcement and call into a study phone line: the study team person king to the individual may obtain non-written consent to ask eligibility questions over the phone. |
| | х | No<br>Yes | <ul> <li>→ If no, skip the rest of this section; go to <u>question 5.1</u>.</li> <li>→ If yes, describe the consent process.</li> </ul> |
| | | | in yes, describe the sonsent processi |
| | | | <ul> <li>a. <u>Documentation of consent</u>. Will you obtain a written or verifiable electronic signature from the subject on a consent form to document consent for all of the <u>recruiting and screening procedures</u>?</li> <li>→ If no, describe the information you will provide during the consent process and for</li> </ul> |
| | | | No which procedures. |
| | | | Yes → If yes, upload the consent form to the <b>Consent Forms and Recruitment Materials</b> page of <b>Zipline</b> . |

### **5 PROCEDURES**

(5.1) Study procedures. Using lay language, provide a complete description of the study procedures, including the sequence, intervention or manipulation (if any), drug dosing information (if any), use of records, time required, and setting/location. If it is available and you think it would be helpful to the IRB: Upload a study flow sheet or table to the Supporting Documents SmartForm in Zipline.

For studies comparing standards of care: It is important to accurately identify the research procedures. See UW IRB <u>POLICY:</u>
<u>Risks of Harm from Standard Care</u> and the draft guidance from the federal Office of Human Research Protections, <u>"Guidance on Disclosing Reasonably Foreseeable Risks in Research Evaluating Standards of Care"; October 20, 2014.</u>

# Aim 1: [redacted]

#### Aim 2:

Once a local health department has been recruited to participate in the study, they will be randomized to one of two conditions for the trial: 1) standard training and technical assistance or 2) standard training plus enhanced technical assistance.

Briefly, local health department staff will be trained to deliver the *Connect to Wellness* intervention to worksites that they recruit. In the Assessment phase, staff will measure current worksite implementation of physical activity, nutrition, cancer screening, and tobacco cessation evidence-based interventions (with the Baseline Employer Assessment Survey). [redacted] At the conclusion of the Implementation phase (month 12), the local health department staff will re-administer the Employer Assessment Survey. After this 12-month period, worksites are able to contact the local health department for technical assistance; the health department may also periodically contact worksites with study updates or to provide relevant materials or offer implementation support.

Once a local health department is assigned to the standard arm, a member of the research team will contact staff to arrange dates for the training sessions, ship materials for the worksites (e.g. toolkits), and provide a detailed *Connect to Wellness* protocol to use with worksites that they recruit. The research team will e-mail information about the *Connect to Wellness* training website and ensure that staff are able to register. Local health department staff will attend three online training webinars, each lasting two hours, in groups of five. (Note: Five refers to the number of local health departments represented in each group). These real-time webinars will be supported by Zoom software. Topics covered in this training will include an introduction to *Connect to Wellness*, methods for recruiting worksites, how to administer the Employer Assessment Survey, how to create and deliver the recommendations report, an overview of intervention implementation and programming, how to track (e.g. their interactions with worksites, time spent on project), and discussion of common barriers and solutions. At the conclusion of the third training webinar, we will work with each group of local health departments to identify a time for monthly group technical assistance calls, where staff will have time to share lessons learned and success stories. Features will be added to the *Connect to Wellness* website to encourage communication between members of each five-local health department group, such as discussion forums and instant chat.

Local health departments assigned to the enhanced arm will undergo initial and online training procedures as described above. Each group will also have a monthly technical assistance call and access to the online peer-communication tools described above. In addition, local health departments in this arm will have one-on-one telephone access to a member of our research team. They can call her for advice; she will proactively contact each local health department in this arm monthly if they have not contacted her during that time. Enhanced support will be given for 24 months, the same length as the study period for this aim.

Throughout the study period, members of the research team will contact local health department staff via e-mail or telephone to obtain study data (measures described in Section 5.2). REDCap will be primarily used for data collection.

Local health department staff will provide members of the research team with the contact information of worksite representatives from a sample of the worksites they recruit and deliver Connect to Wellness to. These representatives will be contacted via e-mail or telephone to schedule a time to complete the brief satisfaction survey. The survey will be administered by telephone.

#### Aim 3:

Following methods recommended by previous studies, we will assess the overall costs to implement the standard and enhanced training and technical assistance strategies, including all training and technical assistance activities conducted by the research team as well as activities performed by local health departments.

(5.2) Data variables. Describe the specific data you will obtain (including a description of the most sensitive items). If you would prefer, you may upload a list of the data variables to the **Supporting Documents** SmartForm instead of describing the variables below.

# Aim 1: [redacted]

#### Aims 2/3:

We will collect the following data from local health department staff: 1) <u>local health department characteristics</u>; 2) <u>satisfaction with training and technical assistance</u>; 3) <u>implementation and intent to maintain *Connect to Wellness*</u>; and 5) <u>staff and worksite activities</u>, which will help us to determine which implementation strategy is more effective and the costs associated with each implementation strategy.

- 1. We will measure local health department characteristics using items from the 2016 National Profile of Local Health Departments. Sample measures include state, population size served, geographic region served, and governance (state, local, or shared). A co-investigator on this grant will pull these measures from the 2016 National Profile data, and we will ask staff to confirm their local health department's information.
- 2. We will ask staff to complete a brief online evaluation to assess satisfaction with and understanding of the training. We will also ask them to complete a satisfaction survey with the *Connect to Wellness* technical assistance they receive every six months and ask staff in the enhanced arm about their satisfaction with one-on-one support.
- 3. We will adapt adoption, implementation, and maintenance items from the Prevention Program Assessment and ask local health department staff to complete these items at 12 and 24 months to assess their implementation and intent to maintain *Connect to Wellness*. The Program Sustainability Assessment Tool will be used as an additional measure to assess capacity to maintain *Connect to Wellness*.
- 4. Staff will be asked to track and provide data on the following: number of meetings, phone contacts, and emails with each worksite; number of worksites that complete *Connect to Wellness*; and personnel time, travel costs, and costs for printing materials for worksites.

In addition to the measures described above, local health department staff will provide us with the Employer Assessment Survey data that they collect from the worksites, which will further help us to determine which implementation strategy is more effective. The identities of the worksite representatives that we ask to complete the brief satisfaction survey will be known to us for recruitment purposes, but we will not retain this information as part of our study data. The identities of these representatives will not be known otherwise. For the employer assessment survey, we will only know the worksite name and corresponding ID number.

Lastly, the research team will track local health department's participation in *Connect to Wellness* training sessions and their attendance at technical assistance calls (group calls and one-on-one calls). The *Connect to Wellness* training and support website will track each local health department's log-ins, visits to the website, and material downloads.

For the worksite representatives, we will collect data on their satisfaction with Connect to Wellness.

5.3) Data sources. For all types of data that you will access or collect for this research: Identify whether you are obtaining the data from the subjects (or subjects' specimens) or whether you are obtaining the data from some other source (and identify the source).

If you have already provided this information in Question 5.1, you do not need to repeat the information here.

Aim 1:

[redacted]

Aims 2/3:

The data described above will come from members of the research team, local health department staff, and worksite representatives.

5.4) Retrospective/prospective. For all types of data and specimens that you will access or collect for this research: do all data and specimens to be used in the research exist (for example, in subjects' medical records) at the time this application is being submitted for initial review?

Yes

No

Include any necessary comments or explanation below (Note that for most studies this can be left blank):

5.5)Identifiability of data and specimens. Answer these questions carefully and completely. This will allow HSD to accurately determine the type of review that is required and to assist you in identifying relevant compliance requirements. Review the following definitions before answering the questions:

Access means to view or perceive data, but not to possess or record it. See, in contrast, the definition of "obtain". Identifiable means that the identity of an individual is or may be readily (1) ascertained by the researcher or any other member of the study team from specific data variables or from a combination of data variables, or (2) associated with the information.

Direct identifiers are direct links between a subject and data/specimens. Examples include (but are not limited to): name, date of birth, medical record number, email or IP address, pathology or surgery accession number, student number, or a collection of your data that is (when taken together) identifiable.

Indirect identifiers are information that links between direct identifiers and data/specimens. Examples: a subject code or pseudonym.

Key refers to a single place where direct identifiers and indirect identifiers are linked together so that, for example, coded data can be identified as relating to a specific person. Example: a master list that contains the data code and the identifiers linked

**Obtain** means to possess or record in any fashion (writing, electronic document, video, email, voice recording, etc.) for research purposes and to retain for any length of time. This is different from accessing, which means to view or perceive data.

a. Will you or any members of your team have access to any direct or indirect identifiers?



→ If yes, describe which identifiers and for which data/specimens.

Aim 1:

[redacted]

Aims 2/3:

We will know the names and contact information of local health department staff and worksite representatives. Electronic data files will refer to all worksites and local health departments via a numerical ID rather than by name.

| No No | → If no, select the reason(s) why you (and all members of your team) will not have access to direct or indirect identifiers. |
|---|---|
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |
| <b>b.</b> Will you <u>obt</u> | ain any direct or indirect identifiers? |
| x Yes | → If yes, describe which identifiers and for which data/specimens. |
| | We have to obtain names and contact information for recruitment and scheduling purposes. |
| No | → If no, select the reason(s) why you (and all members of your team) will not obtain direct or indirect identifiers. |
| | There will be no identifiers. |
| | Identifiers or the key have been (or will have been) destroyed before you have access. |
| | You have (or will have) entered into an agreement with the holder of the identifiers (or key) that prohibits the release of the identifiers (or key) to you under any circumstances. |
| | You should be able to produce this agreement for IRB upon request. Examples: a Data Use Agreement, Repository Gatekeeping form, or documented email. |
| | There are written policies and procedures for the repository/database/data management center that prohibit the release of the identifiers (or identifying link). This includes situations involving an Honest Broker. |
| | There are other legal requirements prohibiting the release of the identifiers or key to you. Describe them below. |
| • | any identifiers, indicate how the identifiers will be stored (and for which data). NOTE: Do not |
| • | any identifiers, indicate how the identifiers will be stored (and for which data). NOTE: Do not are data security plan here – we will ask for that information in section 9.6. You will store the identifiers with the data. Describe the data to which this applies: |

| the | u will store identifiers and study data separately but you will maintain a link between e identifiers and the study data (for example, through the use of a code). Describe the ta to which this applies: |
|---|---|
| Fol | r Aim 1, [redacted] |
| de | e will use ID numbers to link study data with participant and organization (local health partment and worksite) names. The file containing these ID numbers will be stored in a parate location. This applies to all data. |
| | u will store identifiers separately from the study data, with no link between the entifiers and the study data. Describe the data to which this applies: |
| | Will individuals who provide you with coded information or specimens for your research r activities for this research? If yes, identify the activities and provide the name of the n/organization. |
| | not limited to: (1) study, interpretation, or analysis of the data that results from the coded and (2) authorship on presentations or manuscripts related to this work. |
| We do not anticipate sha | aring data with anyone outside the study team. |
| 5.6 Newborn dried blood spots. Wi | ill you use newborn dried bloodspots collected in the United States on or after March |
| x No Yes → If yes, is this rese award that prov | earch supported by any federal funding (including any fellowship or career development ides salary support)? If yes, describe how you will ensure that the bloodspots were collected with parental permission (in compliance with a 2015 law that applies to federal-funded research). |
| reason (for example, to identify | <b>PHI).</b> Will you access, obtain, use, or disclose a participant's identifiable PHI for any or screen potential subjects, to obtain study data or specimens, for study follow-up) on or obtaining of a Limited Data Set? |
| | althcare record information or clinical specimens from an organization considered a "covered ons, in any form or media, whether electronic, paper, or oral. <b>If you will use UW Medical or this question.</b> |
| • | est of this question; go to <u>question <b>5.8</b></u> |
| Yes → If yes, answer a | Il of the questions below. |

| <b>a.</b> Describe the PHI you will access or obtain, and the reason for obtaining it. <i>Be specific</i> . |
|---|
| <b>b.</b> Is any of the PHI located in Washington State? |
| No<br>Yes |
| c. Describe how you will access or obtain the PHI. Be specific. |
| d. For which PHI will you obtain HIPAA authorization from the subjects by having them sign a HIPAA<br>Authorization form, before obtaining and using the PHI? |
| Confirm by checking the box that you will use the UW Medicine HIPAA Authorization form maintained on the HSD website if you will access, obtain, use, or disclose UW Medicine PHI. |
| Confirmed |
| e. For which PHI will you NOT obtain HIPAA authorization from the subjects? |
| Provide the following assurances by checking the boxes. |
| The PHI will not be reused or disclosed to any other person or entity, except as required by law, for authorized oversight of the research study, or for other research for which the use or disclosure of PHI would be permitted. |
| You will fulfill the HIPAA "accounting for disclosures" requirement. See <a href="UW Medicine Privacy">UW Medicine Privacy</a> <a href="Policy #25">Policy #25</a> . THIS IS ONLY FOR UW RECORDS. |
| There will be reasonable safeguards to protect against identifying, directly or indirectly, any patient in any report of the research. |
| 6.8 Genomic data sharing. Will you obtain or generate genomic data (as defined at http://osp.od.nih.gov/scientific-sharing/genomic-data-sharing-faqs/)? |
| x No |
| Yes $\rightarrow$ If yes, answer the question below. |
| a. Do you plan to send genomic data from this research to a national database (for example, NIH's dbGaP database)? |
| No Yes → If yes, complete the <u>ZIPLINE SUPPLEMENT Genomic Data Sharing</u> and upload it to the <b>Supporting Documents</b> SmartForm of <b>Zipline</b> . |

5.9 Whole genome sequencing. For research involving biospecimens: Will the research include whole genome sequencing?

Whole genome sequencing is sequencing of a human germline or somatic specimen with the intent to generate the genome or exome sequence of that specimen.



5.10 Data and specimen sharing/banking. Are you likely to share some or all of the data, specimens, or subject contact information with other researchers or a repository/database for research purposes not related to this study, or to bank them for your own future unspecified research uses? You are strongly encouraged to consider the broadest possible future plans you might have, and whether you will obtain consent now from the subjects for future sharing or unspecified uses. Answer YES even if you will only share information without identifiers. Answer NO if you are unlikely to do any sharing, or if your only sharing will be through the NIH Genomic Data Sharing described in question 5.8.

Many federal grants and contracts now require data or specimen sharing as a condition of funding, and many journals require data sharing as a condition of publication. "Sharing" may include: informal arrangements to share your banked data/specimens with other investigators; establishing a repository from which you formally share with others through written agreements; or sending your data/specimens to a third party repository/archive/entity such as the Social Science Open Access Repository (SSOAR), or the UCLA Ethnomusicology Archive.



→ If yes, answer all of the questions below.

**a.** Describe <u>what will be stored</u>, including whether any direct or indirect (e.g., subject codes) identifiers will be stored.

For Aims 2/3, we will store participant names and contact information (e-mail address, mailing address, and/or telephone number). All participants will be assigned an indirect identifier, so this information will also be stored.

**b.** Describe <u>what will be shared</u>, including whether direct identifiers will be shared and (for specimens) what data will be released with the specimens.

All of the information described above in (a) will be shared.

c. Who will oversee and/or manage the sharing?

A member of the research team will oversee and manage the sharing (e.g. research coordinator).

**d.** Describe the possible future uses, including limitations or restrictions (if any) on future uses or users. As stated above, consider the broadest possible uses.

Examples: data will be used only for cardiovascular research; data will not be used for research on population origins.

The names and contact information may be used to communicate with participants about other research studies related to workplace health promotion and chronic disease prevention (e.g. whether they would be interested in participating).

e. Consent. Will you obtain consent now from subjects for the banking and/or future sharing?



→ If yes, be sure to include the information about this consent process in the consent form (if there is one) and in your answers to the consent questions in Section 8.

f. Withdrawal. Will subjects be able to withdraw their data/specimens from banking or sharing?

No

Yes → If yes, describe how, and whether there are any limitations on withdrawal.

Example: data can be withdrawn from the repository but cannot be retrieved after they are released.

If participants indicate that they do not want to have their information banked

**g.** Agreements for sharing or release. Confirm by checking the box that you will comply with UW (and, if applicable, UW Medicine) policies that require a formal agreement between you and the recipient for release of data or specimens to individuals or entities other than federal databases.

and shared, it will be removed from our records after this study has ended.

Data Use Agreements or Gatekeeping forms are used for data; Material Transfer Agreements are used for specimens (or specimens plus data). Do not attach your template agreement forms; the IRB neither reviews nor approves them

X Confirmed

**5.11 Communication with subjects during the study**. Describe the types of communication (if any) you will have with already-enrolled subjects during the study. Provide a description instead of the actual materials themselves.

Examples: email, texts, phone, or letter reminders about appointments or about returning study materials such as a questionnaire; requests to confirm contact information.

# Aim 1: [redacted]

Aims 2/3:

Research team members will have multiple types of contact with the local health department staff, including emails, phone calls, and in-person meetings. Research team members' only direct contact with worksite representatives will be to collect their brief satisfaction survey data once, after the worksite has been doing Connect to Wellness for 12 months.

**5.12 Future contact with subjects**. Do you plan to retain any contact information you obtain for your subjects so that they can be contacted in the future?

| | No |
|---|----|
| х | Ye |

→ If yes, describe the purpose of the future contact, and whether use of the contact information will be limited to your team; if not, describe who else could be provided with the contact information.

Describe your criteria for approving requests for the information.

Examples: inform subjects about other studies; ask subjects for additional information or medical record access that is not currently part of the study proposed in this application; obtain another sample.

#### Aim 1:

[redacted]

### Aims 2/3:

As mentioned above, participants' name and contact information will be retained. This information may be used to communicate with participants about other research studies related to workplace health promotion and chronic disease prevention.

# **5.13 Alternatives to participation.** Are there any alternative procedures or treatments that might be advantageous to the subjects?

If there are no alternative procedures or treatments, select "No". Examples of advantageous alternatives: earning extra class credit in some time-equivalent way other than research participation; obtaining supportive care or a standard clinical treatment from a health care provider instead of participating in research with an experimental drug.

| х | No |
|---|----|
| | V- |

**Yes** → If yes, describe the alternatives.

- **5.14 Upload to the Supporting Documents** SmartForm of *Zipline* all data collection forms (if any) that will be directly used by or with the subjects, and any scripts/talking points you will use to collect the data. Do not include data collection forms that will be used to abstract data from other sources (such as medical or academic records, or video recordings.
  - **Examples**: survey, questionnaires, subject logs or diaries, focus group questions.
  - NOTE: Sometimes the IRB can approve the general content of surveys and other data collection instruments rather than the specific form itself. This prevents the need to submit a modification request for future minor changes that do not add new topics or increase the sensitivity of the questions. To request this general approval, use the text box below to identify the questionnaires/surveys/ etc. for which you are seeking this more general approval. Then briefly describe the scope of the topics you will cover and the most personal and sensitive questions. The HSD staff person who screens this application will let you know whether this is sufficient or whether you will need to provide more information.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.
  - For data that will be gathered in an evolving way: This refers to data collection/questions that are not pre-determined but rather are shaped during interactions with participants in response to observations and responses made during those interactions. If this applies to your research, provide a description of the process by which you will establish the data collection/questions as you interact with subjects, how you will document your data collection/questions, the topics you plan to address, the most sensitive type of information you will plan to gather, and the limitations (if any) on topics you will raise or pursue.

### Use this text box (if desired) to provide:

- Short written descriptions of materials that cannot be uploaded, such as URLs
- A description of the process you will use for data that will be gathered in an evolving way.
- The general content of questionnaires, surveys and similar instruments for which you are seeking general approval. (See the **NOTE** bullet point in the instructions above.)

| Aim | 1: |
|-----|------------|
| | [redacted] |

**5.15 Send HSD** a <u>Confidentiality Agreement</u> if you will obtain or use any private identifiable UW records without subject's written consent (for example, screening medical records or class grades to identify possible subjects).

The Confidentiality Agreement form must be completed, printed, signed, and mailed to the Human Subjects Division at Box 359470. Your IRB application cannot be approved until we receive the Confidentiality Agreement.

## 6 CHILDREN (MINORS) and PARENTAL PERMISSION

**(6.1)Involvement of minors.** Does your research include minors (children)?

**Minor or child** means someone who has not yet attained the legal age for consent for the research procedures, as described in the applicable laws of the jurisdiction in which the research will be conducted. This may or may not be the same as the definition used by funding agencies such as the National Institutes of Health.

- In Washington State the generic age of consent is 18, meaning that anyone under the age of 18 is considered a child.
- There are some procedures for which the age of consent is much lower in Washington State.
- The generic age of consent may be different in other states, and in other countries.

| x No → If no, go to Section 8. Yes → If we provide the age range of the minor subjects for this study and the legal age for consent in wo | | | | |
|---|---|---|---|---|
| | → If yes, provide the age range of the minor subjects for this study and the legal age for consent in your population(s). If there is more than one answer, explain. | | | |
| | Don't | <ul> <li>→ This means is it not possible to know the age of your subjects. For example, some research involving social media, the Internet, or a dataset that you obtaresearcher or from a government agency. Go to <a href="Section 8">Section 8</a>.</li> </ul> | | |
| as<br>the | <b>5.2 Parental permission. Parental permission</b> means actively obtaining the permission of the parents. This is <u>not</u> the same as "passive" or "opt out" permission where it is assumed that parents are allowing their children to participate because they have been provided with information about the research and have not objected or returned a form indicating they don't want their children to participate. | | | |
| a. | Will you o | obtain parental permission for: | | |
| | All of | your research procedures $\rightarrow$ Go to <u>question 6.2b.</u> | | |
| | None | of your research procedures Use the table below to provide your justification, 6.2b. | and skip o | uestion |
| | Some | of your research procedures Use the table below to identify the procedures for not obtain written parental permission. | or which yo | ou will |
| | | onsider all research procedures and plans, including screening, future contact, and sharing/bai<br>or future work. | nking of da | ta and |
| | nildren<br>Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO parental permission <sup>2</sup> Reason why you will not obtain parental permission | Will you<br>them ab<br>resea | out the |
| | | | YES | NO |

| <ol> <li>If your answer is the same for all children groups or all procedures, you can collapse your answer across procedures.</li> <li>If you plan to obtain identifiable information or biospecimens without parent permission, any waiver g not override parents' refusal to provide broad consent (for example, through the Northwest Biotrust).</li> <li>Will you inform them about the research beforehand even though you are not obtaining active permission</li> <li>b. Indicate by checking the appropriate box(es) your plan for obtaining parental permission</li> <li>Both parents, unless one parent is deceased, unknown, incompetent, or not reasonably arone parent has legal responsibility for the care and custody of the child</li> </ol> | ranted by the | : IRB does |
|---|---|---|
| One parent, even if the other parent is alive, known, competent, reasonably available, and responsibility for the care and custody of the child. | d shares lega | I |
| This is all that is required for minimal risk research. | | |
| If you checked both boxes, explain: | | |
| 6.3 Children who are wards. Will any of the children be wards of the State or any other agency, institution No Yes → If yes, an advocate may need to be appointed for each child who is a ward. The adaddition to any other individual acting on behalf of the child as guardian or in loco individual can serve as advocate for all children who are wards. Describe who will be the advocate(s). Your answer must address the following page 1. Packground and experience. | vocate must<br>parentis. Th | be in |
| <ul> <li>Background and experience</li> <li>Willingness to act in the best interests of the child for the duration of th</li> <li>Independence of the research, research team, and any guardian organize</li> </ul> | | |

## **7 ASSENT OF CHILDREN (MINORS)**

Go to <u>Section 8</u> if your research does not involve children (minors).

**7.1 Assent of children (minors)**. Though children do not have the legal capacity to "consent" to participate in research, they should be involved in the process if they are able to "assent" by having a study explained to them and/or by reading a simple form about the study, and then giving their verbal choice about whether they want to participate. They may also provide a written assent if they are older. See **WORKSHEET: Children** for circumstances in which a child's assent may be unnecessary or inappropriate.

| All of your research | n procedures and child groups | → Go to guestion <b>7.2.</b> |
|---|---|---|
| None of your resea | arch procedures and child groups | <ul> <li>→ Use the table below to provide your justification, then skip to question 7.5.</li> <li>→ Use the table below to identify the procedures for which you will not obtain assent.</li> </ul> |
| Some of your resea | arch procedures and child groups | |
| Be sure to consider all resea<br>specimens for future work. | arch procedures and plans, including screen | ing, future contact, and sharing/banking of data and |
| Children Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which assent will NOT be obtained | Reason why you will not obtain assent |
| | for all children groups or all procedures, you | u can collapse your answer across the groups and/or |
| procedures. | | |
| ages, answer separately fo | • | group. If your research involves children of different glish speakers, include a description of how you will |
| ages, answer separately fo | or each group. If the children are non-Eng | <del>-</del> |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description | or each group. If the children are non-Englend the information you provide. | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Desiverbal indications) during | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object the research, and what you will do in res | glish speakers, include a description of how you will |
| ages, answer separately for ensure that they compreh 7.3 Dissent or resistance. Description of assent. 7.4 Documentation of assent. assent? | or each group. If the children are non-Englend the information you provide. cribe how you will identify a child's object the research, and what you will do in res | glish speakers, include a description of how you will cition or resistance to participation (including non-sponse. |
| ages, answer separately for ensure that they comprehence. 7.3 Dissent or resistance. Deserverbal indications) during 7.4 Documentation of assent. assent? None of your research. | or each group. If the children are non-Engiend the information you provide. cribe how you will identify a child's object the research, and what you will do in research. | glish speakers, include a description of how you will ction or resistance to participation (including non-sponse. ribes whether you will obtain documentation of → Use the table below to provide your |

| | Children | Describe the procedures or data/specimen collection (if any) for which assent |
|---|---|---|
| | Group <sup>1</sup> | will NOT be documented |
| | · | |
| Table | footnotes | |
| 1. If | | ne for all children groups or all procedures, you can collapse your answer across the groups and/or |
| ć | a. Describe how you value a description of wh | will document assent. If the children are functionally illiterate or are not fluent in English, include nat you will do. |
| CI<br>OI<br>OI<br>SU | the information she in Word, if possible hildren who reach the hildren who were enrotain it for the first time hildren who reach the higoing interactions or object's identify is rea | ine. Assent materials are not required to provide all of the standard elements of adult consent; ould be appropriate to the age, population, and research procedures. The documents should be elements age of consent during participation in longitudinal research. Olled at a young age and continue for many years: It is best practice to re-obtain assent (or to me, if you did not at the beginning of their participation). Elegal age of consent: You must obtain informed consent from the now-adult subject for (1) any interventions with the subjects, or (2) the continued analysis of specimens or data for which the dily identifiable to the researcher, unless the IRB waives this requirement. |
| 1 | <ul> <li>If you plan to contact.</li> </ul> | s (if any) to obtain consent for children who reach the legal age of consent. obtain consent, describe what you will do about now-adult subjects whom you are unable to plan to obtain consent or think that you will be unable to do so, explain why. |
| | | rements. (This is for your information only; no answer or response is required.) Researchers are ining whether their research conducted in schools, with student records, or over the Internet |

- comply with permission, consent, and inspection requirements of the following federal regulations:
  - PPRA Protection of Pupil Rights Amendment
  - FERPA Family Education Rights and Privacy Act
  - COPPA Children's Online Privacy Protection Act

## **8 CONSENT OF ADULTS** Review the following definitions before answering the questions in this section. is the process of informing potential subjects about the research and asking them whether they want to participate. It usually (but not always) includes an opportunity **CONSENT** for subjects to ask questions. It does not necessarily include the signing of a consent form. This question is about the consent process. refers to how a subject's decision to participate in the research is documented. This is CONSENT DOCUMENTATION typically obtained by having the subject sign a consent form. is a document signed by subjects, by which they agree to participate in the research as **CONSENT FORM** described in the consent form and in the consent process. are specific information that is required to be provided to subjects. **ELEMENTS OF CONSENT** is the parent's active permission for the child to participate in the research. Parental PARENTAL PERMISSION permission is subject to the same requirements as consent, including written documentation of permission and required elements. is an alternative way of obtaining written documentation of consent that is most SHORT FORM CONSENT commonly used with individuals who are illiterate or whose language is one for which translated consent forms are not available. means there is IRB approval for not obtaining consent or for not including some of the elements of consent in the consent process. **WAIVER OF CONSENT NOTE**: If you plan to obtain identifiable information or identifiable biospecimens without consent, any waiver granted by the IRB does not override a subject's refusal to provide broad consent (for example, the Northwest Biotrust). WAIVER OF DOCUMENTATION means that there is IRB approval for not obtaining written documentation of consent. OF CONSENT **8.1 Groups** Identify the groups to which your answers in this section apply. Adult subjects Parents who are providing permission for their children to participate in research → If you selected **PARENTS**, the word "consent" below should also be interpreted as applying to parental permission and "subjects" should also be interpreted as applying to the parents. 8.2 The consent process. This series of questions is about whether you will obtain consent for all procedures except recruiting and screening and, if yes, how. The issue of consent for recruiting and screening activities is addressed in question 4.6. You do not need to repeat your answer

ZIPLINE APPLICATION: IRB Protocol

a. Are there any procedures for which you will not obtain consent?

| х | No |
|---|----|
| | Ye |

to question 4.6.

→ If yes, use the table below to identify the procedures for which you will not obtain consent. "All" is an acceptable answer for some studies.

Be sure to consider all research procedures and plans, including future contact, and sharing/banking of data and specimens for future work.

| Group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO consent process | Reason why you will not obtain<br>consent | Will<br>prov<br>subject<br>info abo<br>researc<br>they fi | vide<br>ts with<br>out the<br>th after |
|---|---|---|---|---|
| | | | YES | NO |

### Table footnotes

- 1. If your answer is the same for all groups you can collapse your answer across the groups and/or procedures.
  - **b.** <u>Describe the consent process</u>, if you will obtain consent for any or all procedures, for any or all groups. Address groups and procedures separately if the consent processes are different.

Be sure to include:

- The location/setting where consent will be obtained
- Who will obtain consent (refer to positions, roles, or titles, not names).
- Whether/how you will provide an opportunity for questions
- How you will provide an adequate opportunity for the subjects to consider all options

### Aim 1:

[redacted]

#### Aims 2/3:

Local health departments that are interested in participating in the study will receive a written memorandum of understanding (MOU) that outlines the project, the research team's responsibilities, and the local health department's responsibilities. The local health department director and the staff person(s) who will participate in the study will sign the MOU. While not legally binding, a signed MOU provides a written record ensuring that (a) the director understands and supports staff member roles in the study and (b) the local health department staff member understands the scale of the training and *Connect to Wellness* goals. The MOU also documents everything UW will provide in terms of training, materials, and TA. We will consider a local health department enrolled in the study after it returns the signed MOU and one or more of their staff attends the first training session. Local health department staff will also be given an information sheet that outlines their responsibilities and contains additional elements of consent. Worksite representatives will be provided with information about the brief satisfaction survey and asked if they would be willing to participate in the survey. The information sheet

given to LHD staff and worksite representatives will inform participants that their name and contact information will be stored for future research projects.

**c.** <u>Comprehension</u>. Describe how you will ensure or test the subjects' understanding of the information during the consent process.

We will ask participants if they have any questions and if they understand the purpose of the study/study procedures.

**d.** <u>Influence</u>. Does your research involve any subject groups that might find it difficult to say "no" to your research because of the setting or their relationship with you, even if you don't pressure them to participate?

Examples: Student participants being recruited into their teacher's research; patients being recruited into their healthcare provider's research, study team members who are participants; outpatients recruited from an outpatient surgery waiting room just prior to their surgery.



→ If yes, describe what you will do, for each of these subject groups, to reduce any effect of the setting or relationship on their decision.

Examples: a study coordinator will obtain consent instead of the subjects' physician; the researcher will not know which subjects agreed to participate; subjects will have two days to decide after hearing about the study.

**e.** Ongoing process. For research that involves multiple or continued interaction with subjects over time, describe the opportunities (if any) you will give subjects to ask questions or to change their minds about participating.

# Aim 1: [redacted]

Aims 2/3:

The local health department staff will be in regular monthly communication with members of the research team via technical assistance support and will be given opportunities to share their experiences with the study and decline to continue participation, if desired.

**8.3 Written documentation of consent.** Which of the statements below describe whether you will obtain documentation of consent? NOTE: This question does not apply to screening and recruiting procedures which have already been addressed in <u>question 4.6</u>.

Documentation of consent that is obtained electronically is not considered written consent unless it is obtained by a method that allows verification of the individual's signature. In other words, saying "yes" by email is rarely considered to be written documentation of consent

**a.** Are you obtaining written documentation of consent for:

| None of your research procedures | → Use the table below to provide your justification then go to question 8.4. |
|---|---|
| All of your research procedures | → Do not complete the table; go to question 8.4. |
| x Some of your research procedures | → Use the table below to identify the procedures for which you will<br>not obtain written documentation of consent from your adult<br>subjects. |

| Adult subject<br>group <sup>1</sup> | Describe the procedures or data/specimen collection (if any) for which there will be NO documentation of consent | Will<br>provide<br>with a v<br>stater<br>describi<br>resea<br>(optio | them written ment ing the arch |
|---|---|---|---|
| Aim 1: State chronic disease directors | We will conduct telephone interviews. | х | |
| Aim 1: Local health department directors | We will conduct telephone interviews. | х | |
| Aim 1: Local health department staff | We will conduct focus group discussions. | х | |
| Aims 2/3: Local<br>health department<br>staff | We will collect data from staff on their local health department's characteristics; satisfaction with training and technical assistance; implementation and intent to maintain <i>Connect to Wellness</i> ; and staff and worksite activities | х | |
| Aims 2/3: Worksite representatives | We will administer brief satisfaction surveys among a sample of worksites recruited by local health department staff. | x | |
| 8.4 Non-English-speaki fluency or literacy i x No Yes → If ye then to t | ing or -reading adult subjects. Will you enroll adult subjects who do not speak Engin English? es, describe the process you will use to ensure that the oral and written information during the consent process and throughout the study will be in a language reading and (for written materials such as consent forms or questionnaires) at an appending/comprehension level. | lish or who<br>on provided<br>ly underst | o lack<br>I to |
| C<br>E | nterpretation. Describe how you will provide interpretation and when. Also, descr<br>qualifications of the interpreter(s) – for example, background, experience, languag<br>English and in the other language, certification, other credentials, familiarity with telated vocabulary in English and the target language. | e proficien | |
| | <u>Translations</u> . Describe how you will obtain translations of all study materials (not just and how you will ensure that the translations meet the UW IRB's requirement that documents will be linguistically accurate, at an appropriate reading level for the papopulation, and culturally sensitive for the locale in which they will be used. | t translate | - |

- 8.5 Barriers to written documentation of consent. There are many possible barriers to obtaining written documentation of consent. Consider, for example, individuals who are functionally illiterate; do not read English well; or have sensory or motor impairments that may impede the ability to read and sign a consent form.
  - a. Describe your plans (if any) for obtaining written documentation of consent from potential subjects who may have

| • | btaining written documentation of consent for any part of your research. |
|---|---|
| | olutions: Translated consent forms; use of the Short Form consent process; reading the form to the person gn it; excluding individuals who cannot read and understand the consent form. |
| | 3, we will exclude local health departments whose local health department directors and staff cannot inderstand the MOU from the study. Given the study population, we do not anticipate that this will |
| "Blinding" subject x No Yes → | you deliberately withhold information or provide false information to any of the subjects? Note: its to their study group/condition/arm is not considered to be deception. If yes, describe what information and why. Example: you may wish to deceive subjects about the purpose of the study. |
| Г | |
| | No Yes → If yes, describe how you will debrief the subjects. Upload any debriefing materials, including talking points or a script, to the Consent Form and Recruitment Materials SmartForm of Zipline. |
| 8.7 Cognitively imparesearch? | aired adults, and other adults unable to consent. Do you plan to include such individuals in your |
| Examples: individint | luals with Traumatic Brain Injury (TBI) or dementia; individuals who are unconscious, or who are significantly |
| x No | → If no, go to <u>question 8.8</u> . |
| Yes | → If yes, answer the following questions. |
| | a. Rationale. Provide your rationale for including this population in your research. |
| | <b>b.</b> Capacity for consent / decision making capacity. Describe the process you will use to determine whether a cognitively impaired individual is capable of consent decision making with respect to your research protocol and setting. |

| | <b>b.1.</b> If you will have repeated interactions with the impaired subjects over a time period when cognitive capacity could increase or diminish, also describe how (if at all) you will reassess decision-making capacity and obtain consent during that time. |
|---|---|
| c. | <u>Permission (surrogate consent)</u> . If you will include adults who cannot consent for themselves, describe your process for obtaining permission ("surrogate consent") from a legally authorized representative (LAR). |
| | For research conducted in Washington State, see the <b>SOP: Legally Authorized Representative</b> to learn which individuals meet the state definition of "legally authorized representative". |
| d. | Assent. Describe whether assent will be required of all, some, or none of the subjects. If some, indicate which subjects will be required to assent and which will not (and why not). Describe any process you will use to obtain and document assent from the subjects. |
| e. | <u>Dissent or resistance</u> . Describe how you will identify the subject's objection or resistance to participation (including non-verbal) during the research, and what you will do in response. |

- **8.8 Consent-related materials**. Upload to the **Consent Forms and Recruitment Materials** SmartForm of **Zipline** all consent scripts/talking points, consent forms, debriefing statements, Information Statements, Short Form consent forms, parental permission forms, and any other consent-related materials you will use.
  - <u>Translations must be included</u>. However, you are strongly encouraged to wait to provide them until you know that the IRB will approve the English versions.
  - <u>Combination forms</u>: It may be appropriate to combine parental permission with consent, if parents are subjects as well as providing permission for the participation of their children. Similarly, a consent form may be appropriately considered an assent form for older children.
  - For materials that cannot be uploaded: upload screenshots or written descriptions that are sufficient to enable the IRB to understand the types of data that will be collected and the nature of the experience for the participant. You may also provide URLs (website addresses) or written descriptions below. Examples of materials that usually cannot be uploaded: mobile apps; computer-administered test; licensed and restricted standardized tests.

### 9 PRIVACY AND CONFIDENTIALITY

**9.1 Privacy protections.** Describe the steps you will take, if any, to address possible privacy concerns of subjects and potential subjects.

Privacy refers to the sense of being in control of access that others have to ourselves. This can be an issue with respect to recruiting, consenting, sensitivity of the data being collected, and the method of data collection.

Examples:

- Many subjects will feel a violation of privacy if they receive a letter asking them to participate in a study because they
  have \_\_\_\_ medical condition, when their name, contact information, and medical condition were drawn from medical
  records without their consent. Example: the IRB expects that "cold call" recruitment letters will inform the subject
  about how their information was obtained.
- Recruiting subjects immediately prior to a sensitive or invasive procedures (e.g., in an outpatient surgery waiting room) will feel like an invasion of privacy to some individuals.
- Asking subjects about sensitive topics (e.g. details about sexual behavior) may feel like an invasion of privacy to some individuals.

Aim 1: [redacted]

For all aims, data will be stored on a secured server at UW. Files will not be identified by participant name.

**9.2 Identification of individuals in publications and presentations**. Do you plan to use potentially identifiable information about subjects in publications and presentations, or is it possible that individual identities could be inferred from what you plan to publish or present?



- **9.3** State mandatory reporting. Each state has reporting laws that require some types of individuals to report some kinds of abuse, and medical conditions that are under public health surveillance. These include:
  - Child abuse
  - · Abuse, abandonment, neglect, or financial exploitation of a vulnerable adult
  - Sexual assault
  - Serious physical assault
  - Medical conditions subject to mandatory reporting (notification) for public health surveillance

Are you or a member of your research team likely to learn of any of the above events or circumstances while conducting your research **AND** feel obligated to report it to state authorities?

| х | No | |
|---|---|---|
| | Yes | $\rightarrow$ If yes, the UW IRB expects you to inform subjects of this possibility in the consent form or during the |
| | | consent process, unless you provide a rationale for not doing so: |

(9.4) Retention of identifiers and data. Check the box below to indicate your assurance that you will not destroy any identifiers (or links between identifiers and data/specimens) and data that are part of your research records until after the end of the applicable records retention requirements (e.g. Washington State; funding agency or sponsor; Food and Drug Administration) for your research. If you think it is important for your specific study to say something about destruction of identifiers (or links to identifiers) in your consent form, state something like "the link between your identifier and the research data will be destroyed after the records retention period required by state and/or federal law."

This question can be left blank for conversion applications (existing paper applications that are being "converted" into a Zipline application.)

See the "Research Data" sections of the following website for UW Records management for the Washington State research rectords retention schedules that apply in general to the UW (not involving UW Medicine data):

http://f2.washington.edu/fm/recmgt/gs/research?title=R

See the "Research Data and Records" information in Section 8 of this document for the retention schedules for UW Medicine Records: <a href="http://www.uwmedicine.org/about/Documents/UWM-Records-Retention-Schedule-v1.6.pdf">http://www.uwmedicine.org/about/Documents/UWM-Records-Retention-Schedule-v1.6.pdf</a>



**9.5** Certificates of Confidentiality. Are you planning to obtain a federal Certificate of Confidentiality for your research data? *NOTE: Answer "No" if your study is NIH funded, because all NIH-funded studies automatically have a Certificate.* 



- 9.6 Data and specimen security protections. Identify your data classifications and the security protections you will provide, referring to the <u>ZIPLINE GUIDANCE</u>: Data and Security Protections for the minimum requirements for each data classification level. You cannot answer this question without reading this document. Data security protections should not conflict with records retention requirements.
  - **a.** Which level of protections will you apply to your data and specimens? If you will use more than one level, describe which level will apply to which data and which specimens.

Level 1

**b.** Use this space to provide additional information, details, or to describe protections that do not fit into one of the levels. If there are any protections within the level listed in 9.6.a which you will *not* follow, list those here.

All project data will be stored on a secured server.

## **10 RISK / BENEFIT ASSESSMENT**

- **10.1** Anticipated risks. Describe the <u>reasonably foreseeable</u> risks of harm, discomforts, and hazards to the subjects and others of the research procedures. For each harm, discomfort, or hazard:
  - Describe the magnitude, probability, duration, and/or reversibility of the harm, discomfort, or hazard, AND
  - Describe how you will manage or reduce the risks. Do not describe data security protections here, these are already described in Question 9.6.
  - Consider possible physical, psychological, social, legal, and economic harms, including possible negative effects on financial standing, employability, insurability, educational advancement or reputation. For example, a breach of confidentiality might have these effects.
  - Examples of "others": embryo, fetus, or nursing child; family members; a specific group.
  - Do not include the risks of non-research procedures that are already being performed.
  - If the study design specifies that subjects will be assigned to a specific condition or intervention, then the condition or intervention is a research procedure even if it is a standard of care.
  - Examples of mitigation strategies: inclusion/exclusion criteria; applying appropriate data security measures to prevent unauthorized access to individually identifiable data; coding data; taking blood samples to monitor something that indicates drug toxicity.
  - As with all questions on this application, you may refer to uploaded documents.

The only risk associated with the study is a breach of confidentiality. This risk is small because security measures are in place to protect all data. Furthermore, the nature of the data gathered is not sensitive. No additional (e.g. physical) risks to subjects are anticipated. Datasets will use study IDs to further help protect participant confidentiality.

**10.2** Reproductive risks. Are there any risks of the study procedures to men and women (who are subjects, or partner of subjects) related to pregnancy, fertility, lactation or effects on a fetus or neonate?

Examples: direct teratogenic effects; possible germline effects; effects on fertility; effects on a woman's ability to continue a pregnancy; effects on future pregnancies.



 $\rightarrow$  If no go to question 10.3

→ If yes, answer the following questions:

a. Risks. Describe the magnitude, probability, duration and/or reversibility of the risks.

**b. Steps to minimize risk**. Describe the specific steps you will take to minimize the magnitude, probability, or duration of these risks.

Examples: inform the subjects about the risks and how to minimize them; require a pregnancy test before and during the study; require subjects to use contraception; advise subjects about banking of sperm and ova.

If you will require the use of contraception: describe the allowable methods and the time period when contraception must be used.

c. Pregnancy. Describe what you will do if a subject (or a subject's partner) becomes pregnant

For example; will you require the subject to immediately notify you, so that you can discontinue or modify the study procedures, discuss the risks, and/or provide referrals or counseling?

01/12/2018 Version 1.7

| 10.3 Unforeseeable risks | . Are there any research procedures that may have risks that are currently unforeseeable? |
|---|---|
| Example: using a drug | g that hasn't been used before in this subject population. |
| x No | |
| Yes $\rightarrow$ If y | yes, identify the procedures. |
| | e under regional or general anesthesiology. Will any research procedures occur while subjects-<br>general or regional anesthesia, or during the 3 hours preceding general or regional anesthesia |
| (supplied for non-res | |
| x No | |
| Yes $\rightarrow$ If y | yes, check all the boxes that apply. |
| | Administration of any drug for research purposes |
| | Inserting an intra-venous (central or peripheral) or intra-arterial line for research purposes |
| | Obtaining samples of blood, urine, bone marrow or cerebrospinal fluid for research purposes |
| | Obtaining a research sample from tissue or organs that would not otherwise be removed during surgery |
| | Administration of a radio-isotope for research purposes** |
| | Implantation of an experimental device |
| | Other manipulations or procedures performed solely for research purposes (e.g., experimental liver dialysis, experimental brain stimulation) |
| | If you checked any of the boxes: You must provide the name and institutional affiliation of a physician anesthesiologist who is a member of your research team or who will serve as a safety consultant about the interactions between your research procedures and the general or regional anesthesia of the subject-patients. If your procedures will be performed at a UW Medicine facility or affiliate, the anesthesiologist must be a UW faculty member. |
| | ** If you checked the box about radio-isotopes: you are responsible for informing in advance all appropriate clinical personnel (e.g., nurses, technicians, anesthesiologists, surgeons) about the administration and use of the radio-isotope, to ensure that any personal safety issues (e.g., pregnancy) can be appropriately addressed. This is a condition of IRB approval. |
| NIH). If required for | <b>nitoring</b> . A Data and Safety Monitoring Plan (DSMP) is required for clinical trials (as defined by your research, upload your DSMP to the <b>Supporting Documents</b> SmartForm in <b>Zipline</b> . If it is er document you are uploading (for example, a Study Protocol, use the text box below to name the the DSMP. |
| N/A | |

| N/A |
|---|
| <b>10.7 Withdrawal of participants.</b> If applicable, describe the anticipated circumstances under which participants will be withdrawn from the research without their consent. Also, describe any procedures for orderly withdrawal of a participant, regardless of the reason, including whether it will involve partial withdrawal from procedures and any intervention but continued data collection or long-term follow-up. |
| N/A |
| 10.8) Anticipated direct benefits to participants. If there are any direct research-related benefits that some or all individual participants are likely to experience from taking part in the research, describe them below: |
| Do not include benefits to society or others, and do not include subject payment (if any). Examples: medical benefits such as laboratory tests (if subjects receive the results); psychological resources made available to participants; training or education that is provided. |
| Aims 2/3: A potential benefit to local health departments is increased capacity to do worksite wellness activities. Worksites and their workers will potentially benefit from this research by creating healthier environments for their workers. 10.9 Individual subjects findings. a. Is it likely that your research will unintentionally discover a previously unknown condition such as a disease, |
| suicidal intentions, or genetic predisposition? No Yes → If yes, explain whether and how you would share the information with the subject. |
| b. Do you plan to share the individual results of any of your study procedures or findings with the subjects – such a genetic test results, laboratory tests, etc.? |
| You should answer YES if your consent form says anything about sharing individual information with subjects. No Yes → If yes, complete and upload the <u>SUPPLEMENT: Participant Results Sharing</u> to the <u>Supporting</u> Documents SmartForm of <i>Zipline</i> |
| 10.10 Commercial products or patents. Is it possible that a commercial product or patent could result from this study? X No Yes → If yes, describe whether subjects might receive any remuneration/compensation and, if yes, how the |
| amount will be determined. |

## 11 ECONOMIC BURDEN TO PARTICIPANTS

**11.1 Financial responsibility for research-related injuries.** Answer this question only if the lead researcher is <u>not</u> a UW student, staff member, or faculty member whose primary paid appointment is at the UW.

Describe who will be financially responsible for research-related injuries experienced by subjects, and any limitations. Describe the process (if any) by which participants may obtain treatment/compensation.

N/A

11.2 Costs to subjects. Describe any research-related costs for which subjects and/or their health insurance may be responsible (examples might include: CT scan required for research eligibility screening; co-pays; surgical costs when a subject is randomized to a specific procedure; cost of a device; travel and parking expenses that will not be reimbursed).

Aims 2/3:

Local health department staff will be responsible for costs related to travel (e.g. going to meet with a worksite) and printing materials for worksites (e.g. *Connect to Wellness* intervention toolkits).

11.3 Reimbursement for costs. Describe any costs to subjects that will be reimbursed (such as travel expenses).

Aims 2/3:

Local health department staff will not be reimbursed for any costs.

### **12 RESOURCES**

- Faculty Advisor. (For researchers who are students, fellows, or post-docs.) Provide the following information about your faculty advisor.
  - Advisor's name
  - Your relationship with your advisor (for example: graduate advisor; course instructor)
  - Your plans for communication/consultation with your advisor about progress, problems, and changes.

N/A

**12.2 Study team communication**. Describe how you will ensure that each study team member is adequately trained and informed about the research procedures and requirements (including any changes) as well as their research-related duties and functions.

There is no study team.

All of the investigators on the study team have been trained on IRB, and we will ensure that all study staff have up to date training prior to contacting any participants. The study team will meet at least every other week throughout the project. Study materials will be stored on a shared drive to ensure that all members have ready access to the latest protocols, instruments, and other project-related materials.

# 13 OTHER APPROVALS, PERMISSIONS, and REGULATORY ISSUES

**13.1 Other regulatory approvals**. Identify any other regulatory approvals that are required for this research, by checking applicable boxes

Do not attach the approvals unless requested by the IRB.

| | Approval | Research for which this is required |
|---|---|---|
| Radiation | Safety | Procedures involving the use of radioactive materials or an ionizing radiatio producing machine radiation, if they are conducted for research rather than clinical purposes. Approvals need to be attached to the Supporting Documents page in <i>Zipline</i> . |
| Institution | nal Biosafety | Procedures involving the transfer/administration of recombinant DNA, DNA/RNA derived from recombinant DNA, or synthetic DNA. |
| RDRC | | Procedures involving a radioactive drug or biological product that is not approved by the FDA for the research purpose and that is being used witho an IND, for basic science research (not to determine safety and effectiveness or for immediate therapeutic or diagnostic purposes). |
| ESCRO | | Procedures involving the use of some types of human embryonic stem cells |
| school, exter | nal site/organization, fundi | y other approvals or permissions that will be obtained. For example: from a ng agency, employee union, UW Medicine clinical unit. |
| school, exter | nal site/organization, fundi | ng agency, employee union, UW Medicine clinical unit. |
| school, exter Do not attach N/A Financial Cor | nal site/organization, fundi | ng agency, employee union, UW Medicine clinical unit. ons unless requested by the IRB. member of the team have a Financial Conflict of Interest (FCOI) in this |